| Division | • | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | : Reporting and Analysis Plan for Study 204471, A multicentre, open label, single arm, 32-week treatment study in subjects with severe eosinophilic asthma not optimally controlled with current omalizumab treatment who are switched from omalizumab to mepolizumab 100mg subcutaneous (the OSMO study). |
|---|---|---|
| <b>Compound Number</b> | : | SB-240563 |
| Effective Date | : | 08-MAY-2017 |

# **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report (CSR) for Protocol 204471.
- The critical components RAP was completed on the 10<sup>th</sup> February 2016. This document represents the final RAP and will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

## **Author's Name and Functional Area:**

| PPD | | 03-MAY-2017 |
|------------------|-------------------------------|--------------|
| Statistician, RD | PCPS QSci Clinical Statistics | 03-WA 1-2017 |

## Agreed by core RAP team (via email):

| PPD | (Project Physician Lead, Respiratory Therapeutic Unit) |
|-----|---------------------------------------------------------------|
| PPD | (Global Medical Affairs Lead, Respiratory Franchise) |
| PPD | (Clinical Investigation Leader, Respiratory Therapeutic Unit) |
| PPD | (Medical Director, Safety Evaluation & Risk Management) |
| PPD | (Manager, Clinical Programming) |

## Approved by:

| PPD | | 08-MAY-2017 |
|--------------|-------------------------------|----------------|
| Director, RD | PCPS QSci Clinical Statistics | U8-IVIA 1-201/ |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | REPO | RTING & | ANALYSIS PLAN SYNPOSIS | 4 |
| 2. | SUMM | MARY OF | KEY PROTOCOL INFORMATION | 6 |
| | 2.1. | | s to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | | ojectives and Endpoints | |
| | 2.3. | Study De | esign | 9 |
| | 2.4. | | al Hypotheses | |
| 3. | PLANI | NED ANA | LYSES | 10 |
| | 3.1. | Interim A | nalyses | 10 |
| | 3.2. | Final Ana | alyses | 10 |
| 4. | ANAL' | YSIS POF | PULATIONS | 11 |
| | 4.1. | Protocol | Deviations | 11 |
| 5. | | | ONS FOR DATA ANALYSES AND DATA HANDLING | 40 |
| | CONV | ENTIONS | S | 12 |
| 6. | STUD | Y POPUL | ATION ANALYSES | 13 |
| | 6.1. | Overviev | v of Planned Analyses | 13 |
| 7. | PRIMA | ARY STAT | FISTICAL ANALYSES | 15 |
| | 7.1. | | Analyses | |
| | | 7.1.1. | Overview of Planned Efficacy Analyses | 15 |
| | | 7.1.2. | Planned Efficacy Statistical Analyses | 16 |
| | | 7.1.3. | Analysis Comparing Against A Historical Placebo Effect | 17 |
| 8. | SECO | NDARY S | STATISTICAL ANALYSES | 18 |
| | 8.1 | Efficacy. | Analyses | 18 |
| | | 8.1.1. | Overview of Planned Efficacy Analyses | 18 |
| | | 8.1.2. | Secondary Efficacy Statistical Analyses | <mark>20</mark> |
| | 8.2. | Safety A | nalyses | 24 |
| | | 8.2.1. | Overview of Planned Analyses | |
| | | 8.2.2. | Adverse Events of Special Interest | |
| | | 8.2.3. | Overview of Planned Clinical Laboratory Analyses | 26 |
| | | 8.2.4. | Overview of Planned Other Safety Analyses | <mark>27</mark> |
| | | | 8.2.4.1. Immunogenicity | 28 |
| 9. | REFE | RENCES. | | 30 |
| 10. | APPE | NDICES | | 31 |
| ٠. | 10.1. | Appendi | x 1: Protocol Deviation Management and Definitions for Per | |
| | | | Population | |
| | 40.0 | 10.1.1. | Exclusions from Per Protocol Population | 32 |
| | 10.2. | | x 2: Time & Events | |
| | 40.0 | | Protocol Defined Time & Events | |
| | 10.3. | | x 3: Assessment Windows & Visit Slotting | |
| | | | Assessment Windows | |
| | | 10.3.2. | Early Withdrawal / Treatment Discontinuation Visits | <b>5</b> / |

| | 10.3.3. Unscheduled Visits | 37 |
|--------|--------------------------------------------------------------|----|
| 10.4. | Appendix 4: Treatment Phases | |
| | 10.4.1. Treatment Phases (Exacerbations) | |
| | 10.4.2. Treatment Phases (Visit Based Efficacy Data) | |
| | 10.4.3. Treatment Phases (Adverse Events) | |
| | 10.4.3.1. Adverse Event Data Derivations | 39 |
| | 10.4.4. Treatment Phases (Concomitant Medications) | |
| 10.5. | Appendix 5: Data Display Standards & Handling Conventions | |
| | 10.5.1. Study Treatment & Subgroup Display Descriptors | 41 |
| | 10.5.2. Baseline Definition & Derivations | |
| | 10.5.2.1. Baseline Definition | |
| | 10.5.2.2. Derivations and Handling of Missing Baseline | |
| | Data | 41 |
| | 10.5.3. Reporting Process & Standards | 41 |
| 10.6. | Appendix 6: Derived and Transformed Data | |
| | 10.6.1. General | |
| | 10.6.2. Study Population | |
| | 10.6.3. Efficacy | |
| | 10.6.4. Safety | |
| 10.7. | Appendix 7: Premature Withdrawals & Handling of Missing Data | |
| 10.7. | 10.7.1. Premature Withdrawals | |
| | 10.7.2. Handling of Missing Data | |
| | 10.7.2.1. Handling of Missing or Partial Dates | |
| 10.8. | Appendix 8: Values of Potential Clinical Importance | |
| 10.0. | 10.8.1. Laboratory Values | |
| 10.9. | Appendix 9: Multicenter Studies | |
| 10.0. | 10.9.1. Methods for Handling Centres | |
| 10 10 | Appendix 10: Examination of Covariates and Subgroups | |
| | 10.10.1. Handling of Covariates | |
| | 10.10.2. Handling of Subgroups | |
| 10.11. | Appendix 11: Model Checking and Diagnostics for Statistical | |
| . • | Analyses | 55 |
| | 10.11.1. Statistical Analysis Assumptions | |
| 10.12. | Appendix 12: Abbreviations & Trade Marks | |
| | 10.12.1. Abbreviations | |
| | 10.12.2. Trademarks | |
| 10.13. | Appendix 13: List of Data Displays | |
| | 10.13.1. Data Display Numbering | |
| | 10.13.1.1. Study Population Tables | |
| | 10.13.1.2. Study Population Figures | |
| | 10.13.1.3. Efficacy Tables | |
| | 10.13.1.4. Efficacy Figures | |
| | 10.13.1.5. Safety Tables | |
| | 10.13.1.6. Safety Figures | |
| | 10.13.1.7. ICH Listings | |
| 10 14 | Appendix 14: Example Mock Shells for Data Displays | |
| | pp = | |

# 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | <ul> <li>This reporting and analysis plan (RAP) details all planned analyses and outputs<br/>required for the final Clinical Study Report (CSR) of study 204471.</li> </ul> |
| | The critical components RAP was completed on the 10 <sup>th</sup> February 2016. This |
| | document represents the final RAP and will be provided to the study team |
| | members to convey the content of the Statistical Analysis Complete (SAC) deliverable. |
| Protocol | This RAP is based on protocol amendment 1 (Dated: 23-MAR-2016) for study 204471 (GSK Document No.: 2015N243304_01) and the latest version of the electronic Case Report Form (eCRF) [eCRF Version 2.1]. |
| Primary | To determine in a pragmatic setting whether there is an improvement in asthma |
| Objective | control, from the beginning to the end of the study, when directly switched from |
| | omalizumab to mepolizumab in subjects with a severe eosinophilic asthma phenotype not optimally controlled on omalizumab. |
| Primary | Mean change from baseline in ACQ-5 score at Week 32 |
| Endpoint | moan onango nom sassimo myto Q o sosto at trook oz |
| Study<br>Design | An open label, single arm, 32-week treatment, multi-center study in subjects with severe eosinophilic asthma not optimally controlled with current omalizumab treatment who are switched from omalizumab to mepolizumab 100mg |
| | administered subcutaneously (SC) every 4 weeks. |
| | Approximately 120 subjects are expected to be treated with open label |
| | mepolizumab. |
| Planned | No interim analysis of data is planned for this study. |
| Analyses | <ul> <li>A complete analysis in accordance with all study objectives and endpoints will be<br/>performed after all subjects have completed the study.</li> </ul> |
| | <ul> <li>Decisions regarding the analyses, specified in this RAP document, will be made<br/>prior to Database Freeze of the study data.</li> </ul> |
| Analysis | The 'All Subjects Enrolled' population will be used to summarise Screen and run- |
| Populations | in failures. |
| | The 'Intent-to-Treat' population will be used as the primary population to |
| | summarise the study population, and to evaluate efficacy, safety and PD/Biomarkers. |
| | The 'Per Protocol' population will also be used as a supporting population to |
| | evaluate efficacy. Subjects excluded will have protocol deviations considered to |
| Hypothesis | <ul> <li>potentially have an effect on efficacy.</li> <li>As there is no control arm within this study, comparisons in ACQ score will be</li> </ul> |
| 11, 20110010 | made back to baseline. |
| | The potential of a 'placebo effect' within the mepolizumab treated subjects was |
| | considered when the study was designed and was estimated as an improvement |
| | of -0.55 from baseline in ACQ score, based on placebo subjects within historical |
| | mepolizumab severe asthma studies. However, when only previous Xolair users were considered, an improvement of -0.11 from baseline in ACQ score was |
| | observed. |
| | This study is designed to test the superiority of mepolizumab 100 mg SC |

| Overview | Key Elements of the RAP |
|---|---|
| | treatment vs. baseline. Improvements will also be assessed against the historical 'placebo effects' estimated from previous mepolizumab studies. Significance tests will be performed at the two-sided 5% alpha level (one-sided 2.5%). |
| Primary<br>Analyses | ACQ-5 score will be analysed using a mixed models repeated measures analyses allowing for covariates of region, use of baseline maintenance oral corticosteroids therapy (OCS vs no OCS), exacerbations in the year prior to the study (as an ordinal variable), and visit (including baseline visit). |
| Secondary<br>Analyses | <ul> <li>SGRQ score will be analysed using a mixed models repeated measures analysis as for ACQ-5.</li> <li>Frequency of clinically significant asthma exacerbations will be analysed using a negative binomial regression analysis</li> <li>Blood eosinophil count will be analysed using a mixed model repeated measures analysis after log transformation</li> </ul> |
| Safety<br>Analysis | Safety data including adverse events, vital signs, clinical laboratory, electrocardiogram (ECG), and immunogenicity data will be summarised descriptively. |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Statistical analysis changes to the originally planned statistical analysis specified in the protocol amendment 1 (Dated: 23-MAR-2016) (GSK Document No.: 2015N243304\_01) are outlined in Table 1.

Table 1 Changes to Protocol Defined Statistical Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rational for Changes |
| Analysis of change from baseline in ACQ, SQRQ scores will be performed using a mixed models repeated measures (MMRM) analysis, allowing for covariates of baseline ACQ score, region, baseline maintenance OCS therapy, exacerbations in the year prior to the study (as an ordinal variable), visit and an interaction term for visit by baseline ACQ score. | Baseline values will be included as a data point in the analysis, and there will be no covariate adjustment made in the model. The change from the baseline at Visit X will be calculated by: Estimated Score at Visit X minus Estimated Score at Baseline. | This is a single treatment arm study and comparisons are being made directly to the baseline values. |
| Clinically significant exacerbations will be analyzed using a generalized linear model with covariates for region, baseline maintenance OCS therapy and number of exacerbations in the year prior to the study (as an ordinal variable). | Clinically significant exacerbations will be examined using a generalized estimating equation (GEE) with no adjustments for covariates. | Generalised estimating equations (GEEs) will compare the on-treatment exacerbation rate to the rate within the 12 months prior to study. |

# 2.2. Study Objectives and Endpoints

The below objectives and endpoints will be assessed when subjects with a severe eosinophilic asthma phenotype who are not optimally controlled on omalizumab are directly switched from omalizumab to mepolizumab:

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To describe in a pragmatic<br>situation/setting whether there is<br>an improvement in asthma<br>control from the beginning to the<br>end of the study | Mean change from baseline in Asthma Control<br>Questionnaire-5 (ACQ-5) score at Week 32 |
| Secondary Objectives | Secondary Endpoints |
| To determine whether there is an improvement in Health related Quality of Life (HR-QoL) | <ul> <li>Mean change from baseline in St. George's<br/>Respiratory Questionnaire (SGRQ) score at Week 32</li> </ul> |
| To determine the frequency of asthma exacerbations | Frequency of clinically significant asthma exacerbations over 32 week treatment |
| To evaluate the pharmacodynamic effects | Ratio to baseline in blood eosinophils at Week 32 |
| Other Objectives | Other Endpoints |
| To determine the response to asthma clinical parameters | <ul> <li>Percentage of subjects achieving a 0.5-point or greater reduction from baseline in ACQ-5 score at Week 32</li> <li>Percentage of subjects achieving a 4-point or greater reduction from baseline in SGRQ score at Week 32</li> <li>Mean change from baseline in pre- and post bronchodilator FEV1 at Week 32</li> <li>Frequency of exacerbations requiring ED visit/hospitalization during the treatment period</li> <li>Subject/Clinician rated response to therapy</li> <li>Mean change from baseline in treatment satisfaction questionnaire</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| <ul> <li>To determine the effect on inflammatory biomarkers</li> <li>To characterize patient treatment</li> </ul> | <ul> <li>Change from baseline in some inflammatory<br/>biomarkers expression at week 32</li> <li>Subject Exit Interviews</li> </ul> |
| benefit of mepolizumab | Safaty Endnainta |
| Safety Objectives To determine the safety, | Safety Endpoints |
| To determine the safety, immunogenicity and tolerability of mepolizumab | <ul> <li>Incidence and frequency of Adverse/Serious Adverse Events (including systemic and injection site reactions)</li> <li>Clinically significant change in electrocardiogram (ECGs)</li> <li>Clinically significant change in vital signs</li> </ul> |

## CONFIDENTIAL

204471

| Objectives | Endpoints |
|------------|-----------------------------|
| | Incidence of immunogenicity |

# 2.3. Study Design

| Overview of S | Study Design a | nd Key | Feature | S | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| omalii | zumab | ersi te | ·h to my | polizun | vah 100 | ma SC a | varud u | iooks | $\neg$ |
| | 1-4 weeks | SVVICE | .11 (0 111) | ponzun | 100 100 | ilig ac e | very 4 v | reens | |
| G-2 WEEKY | 1-4 Weeks | | | | | | | | _ |
| | <u> </u> | <u> </u> | | | | | | 120 | 915 |
| V0 V. | l V2<br>(baseline<br>Week 0 | V3<br>) W4 | ∨4<br>∨∨8 | V5<br>W12 | V6<br>W16 | V7<br>VV20 | V8<br>VV24 | ∨9<br>\∀28 | ∀10<br>₩32 |
| Design<br>Features | <ul> <li>An open with seve omalizum 100mg at are not o through t ≥1.5 and</li> </ul> | re eosing<br>ab treatr<br>dminister<br>with seven<br>otimally one ACQ- | ophilic ament whed subcere eosing controllers with a | sthma no<br>o are swi<br>utaneous<br>ophilic as<br>d will be<br>screenin | t optimal<br>tched fro<br>sly (SC) e<br>sthma wl<br>eligible to<br>g (Visit 1 | lly contro<br>om omali<br>every 4 w<br>ho are re<br>o particip<br>) and ba | olled with<br>zumab to<br>veeks.<br>eceiving o<br>eate and v<br>seline (V | current<br>o mepoliz<br>omalizum<br>will be ide<br>isit 2) sco | umab<br>ab, but<br>entified |
| Dosing | period, in<br>Omalizur<br>SC) ever<br>therapies | cluding (<br>nab treat<br>/ 4 week<br>). If patie | Omalizur<br>ment an<br>s for 32<br>ents requ | nab. At V<br>d be swit<br>weeks (tl<br>iire any a | risit 2 sul<br>ched to onere is no<br>dditional | bjects wi<br>open-lab<br>o wash-c<br>mainten | Il discont<br>el mepoli<br>out perioc<br>ance the | inue their<br>izumab (*<br>d betweer<br>rapy (exc | 100 mg<br>n the<br>cept for |
| Treatment<br>Assignment | | | | | | | | | |
| Planned<br>Analysis | <ul> <li>No interir</li> <li>A complete be performed.</li> <li>Decisionse made priorities.</li> </ul> | te analys<br>med afte<br>regardii | sis in acc<br>r all subj<br>ng the al | cordance<br>jects hav<br>nalyses, | with all se comple<br>specified | study objected the states in this F | jectives a<br>study. | · | |

# 2.4. Statistical Hypotheses

This study is designed to investigate whether subjects not optimally controlled on omalizumab can be effectively and safely switched to treatment with mepolizumab to improve asthma control. As there is no control arm in this study, comparisons in ACQ-5 score will be made to baseline. The first hypothesis to be tested will be for superiority of mepolizumab 100 mg SC treatment vs. baseline.

The potential of a 'placebo effect' within the mepolizumab treated subjects has been considered. In the protocol this was estimated as an improvement of -0.55 (SE: 0.05) from baseline in ACQ-5 score, based on the placebo effect observed in mepolizumab subjects from Phase 3 severe asthma studies (meta-analysis of double-blind studies MEA112997 and MEA115588). Improvements from baseline in ACQ-5 score will be assessed against this historical 'placebo effect'. For further information regarding this historical 'placebo effect' please refer to Section 7.1.3.

Significance tests will be performed at the two-sided 5% alpha level (one-sided 2.5%).

## 3. PLANNED ANALYSES

## 3.1. Interim Analyses

No interim analysis of data is planned for this study.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects<br>Enrolled (ASE)<br>Population | Comprised of all subjects enrolled and for whom a record exists on the study database. | Screen and run-in failures |
| Intent-to-Treat<br>(ITT) Population | Comprised of all subjects who receive at least one dose of mepolizumab. | <ul><li>Study Population</li><li>Efficacy</li><li>Safety</li></ul> |
| Per Protocol (PP)<br>Population | Comprised of all subjects in the ITT population who have not been identified as full protocol deviators with respect to criteria that are considered to impact the primary efficacy analysis. The decision to exclude a subject from the PP Population or exclude part of their data from the PP Population analyses will be made prior to freezing the study database. Protocol deviations that would exclude subjects from the PP population are defined in Section 4.1 (Protocol Deviations) and (Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population). | Supplementary analysis of the primary endpoint |

#### NOTES:

 Please refer to Appendix 13: List of Data Displays which details the population to be used for each displays being generated.

#### 4.1. Protocol Deviations

- All protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the Per Protocol analysis are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Important deviations which result in exclusion from the Per Protocol population will also be summarised and listed. (Please refer to Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population).
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 2 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 2 Overview of Appendices

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| 10.2 | Appendix 2: Time & Events |
| 10.3 | Appendix 3: Assessment Windows & Visit Slotting |
| 10.4 | Appendix 4: Treatment Phases |
| 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 10.6 | Appendix 6: Derived and Transformed Data |
| 10.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| 10.8 | Appendix 8: Values of Potential Clinical Importance |
| 10.9 | Appendix 9: Multicenter Studies |
| 10.10 | Appendix 10: Examination of Covariates and Subgroups |
| 10.11 | Appendix 11: Model Checking and Diagnostics for Statistical Analyses |
| Other RA | P Appendices |
| 10.12 | Appendix 12: Abbreviations & Trade Marks |
| 10.13 | Appendix 13: List of Data Displays |
| 10.14 | Appendix 14: Example Mock Shells for Data Displays |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population analyses will be based on the Intent-To-Treat (ITT) population, unless otherwise specified.

Table 3 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 13: List of Data Displays.

 Table 3
 Overview of Planned Study Population Analyses

| Endpoint / Parameter / Display Type | Data Displays Generated | | |
|---|---|---|---|
| | Table | Figure | Listing |
| Subject Disposition | | | |
| Analysis Populations | Υ | | |
| Reasons for Screen and Run-in Failure | Υ | | Y |
| Failed Inclusion/Exclusion/Continuation criteria | Υ | | Υ |
| Subjects by Region, Country and Site | Υ | | |
| Reasons for Subject Withdrawal From Study | Υ | | Y |
| Reasons for Subject Withdrawal From Investigational Product | Υ | | Y |
| Time to Withdrawal From Investigational Product | | <b>Y</b> [1] | |
| Demographic and Baseline Characteristics | | | |
| Demographic Characteristics | Y | | Υ |
| Age Ranges | Y | | |
| Race and Racial Combinations | Υ | | <b>Y</b> [2] |
| Race and Racial Combination Details | Υ | | |
| Demographic and Baseline Disease Characteristics | | | |
| Asthma History and Baseline Disease Characteristics | Y | | |
| Previous Exacerbation History | Y | | |
| History of Tobacco Use | Υ | | |
| Baseline Lung Function Results | Υ | | |
| Past and Current Medical Conditions | Υ | | |
| Cardiovascular Assessments (Family History/Screen Questions) | Υ | | |
| Prior and Concomitant Medications | | | |
| History Xolair Use (including regime, duration of treatment) | Υ | | |
| Asthma Concomitant Medications by Respiratory Medication Class | Y | | |
| Non-Asthma Concomitant Medications Taken During Treatment | Υ | | |
| Relationship between ATC level 1, Ingredient and verbatim text | | | Y |

| Endpoint / Parameter / Display Type | Data Displays Generated | | |
|---|---|---|---|
| | Table | Figure | Listing |
| Protocol Deviations | | | |
| Important Protocol Deviations | Υ | | Υ |
| Protocol Deviations Resulting in Exclusion from PP Population | | | Y |

NOTES: Y = Yes display generated. [1] Kaplan Meier plot; [2] Listing of race as collected in eCRF.

# 7. PRIMARY STATISTICAL ANALYSES

# 7.1. Efficacy Analyses

# 7.1.1. Overview of Planned Efficacy Analyses

The primary efficacy analyses will be based on the Intent-To-Treat (ITT) population. Additional sensitivity analysis will be performed on the Per Protocol population.

Table 4 provides an overview of the planned efficacy analyses, with full details of data displays being presented in Appendix 13: List of Data Displays.

Table 4 Overview of Planned Efficacy Analyses

| Endpoint | | Absolute [1] | | | | | Change from Baseline [1] | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats Analysis | | Sum | mary | Individual | | Stats Analysis | | Summary | | Individual | | | |
| | Т | F | L | T | F | F | L | T | F | L | T | F | F | L |
| Primary Endpoint | | | | | | | | | | | | | | |
| <b>Asthma Control Questi</b> | onnai | re (AC | CQ-5) | | | | | | | | | | | |
| On-treatment & Off- | Y <sup>[4]</sup> | | | Υ | | | | Y <sup>[4]</sup> | <b>Y</b> [5] | | Υ | Υ | | Υ |
| treatment [2] [3] | | | | | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Absolute and change from baseline summaries combined into a single display.
- 2. To be generated for Intent-To-Treat (ITT) population and Per-Protocol (PP) population.
- 3. Subgroup analyses to be repeated for Intent-To-Treat (ITT) population and all subgroups listed within Section
- 4. Table to include both Least Square Means and Least Square Mean Changes and estimated treatment difference (Mepolizumab-Historical Placebo) and 95% confidence interval at each visit from Mixed Model Repeated Measures (MMRM) Analysis.
- 5. Figure to present Least Square Mean Changes and corresponding 95% confidence intervals at each visit from MMRM Analysis

#### 7.1.2. Planned Efficacy Statistical Analyses

## **Primary Statistical Analyses**

## Endpoint(s)

Mean change from baseline in ACQ-5 score at Week 32 (ADaM Dataset : ADACQ5)

#### **Model Specification**

- Endpoint will be analysed using a mixed models repeated measures (MMRM) analysis
- Dependent variable will be ACQ-5 score at each visit including the baseline
- Terms fitted in the MMRM analysis will include:

Fixed Categorical Covariates: Region, Baseline maintenance OCS use, Visit

Fixed Continuous Covariates: Exacerbations in the year prior to study (as an ordinal

variable),

Repeated: Visit

See Section 10.10.1 for further details around model covariates.

# **Model Checking & Diagnostics**

Refer to Appendix 11: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Adjusted means and the corresponding 95% confidence intervals will be presented by visit.
- The estimated adjusted means will be presented using the observed marginal distribution of the sample covariates (OM option in LSMEANS statement).
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used (DDMF=KR).
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line.
- Change from the baseline at each Visit X will be calculated by (Estimated Score at Visit X minus Estimated Score at Baseline) and the corresponding 95% confidence intervals.
   Adjusted means at each visit will also be presented.
- Plots of LS means change from baseline in ACQ-5 Score and 95% confidence intervals from the model will be generated by visit.
- Adjusted mean and corresponding standard error of mean will be presented, together with estimated between treatment difference (Mepolizumab – Historical Placebo) and the corresponding 95% confidence intervals at Week 32.

#### **Treatment Phase**

- All subjects in the ITT population will be included within this analysis.
- All data collected up to and including Week 32 from patients, including those who have discontinued study treatment, will be included in the analysis.

#### **Sensitivity and Supportive Statistical Analyses**

- Additional comparisons to historical placebo effect will be presented at Week 32 (refer to Section 7.1.3 for more details).
- A supporting sensitivity analysis of the Per Protocol (PP) population will also be performed.
- Subgroup analyses of the primary endpoint will be performed for all subgroups listed within Section 10.10.2.

## 7.1.3. Analysis Comparing Against A Historical Placebo Effect

We will perform two separate analyses of the primary endpoint comparing to a historical 'placebo effect'.

Firstly, as specified in the protocol, a meta-analysis of previous exacerbation double-blind studies, MEA112997 and MEA115588, gave an estimate of -0.55 (SE: 0.05), for the improvement in the ACQ-5 score for placebo subjects at Week 32 compared to baseline. The observed improvement in this study for following mepolizumab treatment will be compared to this historical improvement on placebo.

Secondly, a meta-analysis has been performed of subjects within studies MEA115588 and 200862 who reported previous Xolair use, which may represent a more comparable population for this study. Study 200862 has completed since the protocol was finalised and previous Xolair usage was not collected in study MEA112997.

At Week 32 an estimate of -0.29 (SE: 0.248) was reported in the MEA115588 study while at Week 24 study 200862 reported an estimate of -0.03 (SE: 0.164) for the improvement in the ACQ-5 score for placebo subjects who previously used Xolair.

Weighted meta-analysis was performed on these values to get the combined estimate of -0.11 (SE: 0.14) for the historical placebo effect (Figure 1). This shows a reduction in the ACQ-5 score, but not as large as that specified in the protocol. The observed improvement in this study for mepolizumab vs. baseline will be also compared to this historical improvement on placebo.





# 8. SECONDARY STATISTICAL ANALYSES

# 8.1 Efficacy Analyses

# 8.1.1. Overview of Planned Efficacy Analyses

The secondary efficacy analyses will be based on the Intent-To-Treat (ITT) population, unless otherwise specified in Appendix 13: List of Data Displays.

Table 5 provides an overview of the planned efficacy analyses, with further details of data displays being presented in Appendix 13: List of Data Displays.

Table 5 Overview of Planned Efficacy Analyses

| Endpoint | | | Α | bsolut | e <sup>[1]</sup> | | | Change from Baseline [1] [2] | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats | Anal | ysis | Sum | mary | Indi | vidual | Stat | ts Ana | alysis | Sum | mary | Indiv | ridual |
| | T | F | L | Т | F | F | Ш | Т | F | L | Т | F | F | L |
| Secondary Endpoints | | | | | | | | | | | | | | |
| St George's Respirato | ory Qu | estio | nnair | e (SGR | (Q) | | | | | | | | | |
| On-treatment & Off- | Υ | | | Υ | | | | Υ | Υ | | Υ | Υ | | |
| treatment | | | | | | | | | | | | | | |
| Blood Eosinophil Cou | | | | 1 | 1 | 1 | | 1 | 1 | | ı | ı | 1 | 1 |
| On-treatment & Off- | Υ | | | Υ | | | | Υ | Υ | | Υ | | | |
| treatment | | | | | | | | | | | | | | |
| On-treatment [3] | Υ | | | | | | | Υ | | | | | | |
| Other Endpoints | | | | | | | | | | | | | | |
| >= 0.5-point reduction | on fro | m ba | selin | e in A | CQ-5 | score | at We | eek 3 | 32 | | | | | |
| On-treatment & Off- | | | | | | | | | | | Υ | Υ | | |
| treatment | | | | | | | | | | | | | | |
| >= 4-point or greate | r redu | ctior | <u>fror</u> | n base | eline ir | ı SG | RQ To | tal s | core | at We | ek 32 | 2 | | |
| On-treatment & Off- | | | | | | | | | | | Υ | Υ | | |
| treatment | | | | | | | | | | | | | | |
| Pre-Bronchodilator | FEV1 | | | | | | | | | | | | | |
| On-treatment & Off- | Υ | | | Υ | | | | Υ | Υ | | Υ | | | |
| treatment | | | | | | | | | | | | | | |
| Post-Bronchodilato | r FEV | 1 | | | | | | | | | | | | |
| On-treatment & Off- | Υ | | | Υ | | | | Υ | Υ | | Υ | | | |
| treatment | | | | | | | | | | | | | | |
| Subject/Clinician Ra | ated R | espo | nse | to The | rapy | | | | | | | | | |
| On-treatment [3] | | | | Υ | | | | | | | | | | |
| <b>Treatment Satisfact</b> | ion Qu | ıesti | onna | ire for | Medic | catio | n (TSC | (M-9) | ) | | | | | |
| On-treatment [3] | | | | Υ | | | | | | | Υ | | | |
| Biomarkers | | | | | | | | | • | | | | | • |
| On-treatment | | | | Υ | | | | | | | Υ | | | |

| Endpoint | | Incidence of Events | | | | | |
|---|---|---|---|---|---|---|---|
| | S | tats Analysi | S | Sum | mary | Individual | |
| | T | F | L | T | F | F | L |
| Secondary Endpoints | | | | | | | |
| Clinically Significant Exacerbations | | | | | | | |
| On-treatment & Off- | <b>Y</b> [4] | | | Υ | Υ | | Υ |
| treatment | | | | | | | |
| On-treatment [3] | <b>Y</b> [4] | | | | | | |
| <b>Exacerbations requir</b> | ing ED visi | it/hospitali | ization | | | | |
| On-treatment & Off- | <b>Y</b> [4] | | | Υ | | | Υ |
| treatment | | | | | | | |
| On-treatment [3] | <b>Y</b> [4] | | | | | | |
| <b>Exacerbations requir</b> | ing hospita | alization | | | | | |
| On-treatment & Off- | Y[4] | | | Υ | | | Υ |
| treatment | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Absolute and change from baseline summaries combined into a single display.
- 2. Ratio to Baseline to be shown for Blood Eosinophil Count and Biomarker data.
- 3. To analyse data collected whilst On-Treatment, not considering any data collected following treatment discontinuation (see Section 10.4).
- 4. Table to include annualised exacerbation rate and 95% confidence intervals from negative binomial model.

## 8.1.2. Secondary Efficacy Statistical Analyses

#### **Secondary Statistical Analyses**

#### Secondary Endpoint(s)

Mean change from baseline in SGRQ at Week 32

# **Model Specification**

See Primary Efficacy Statistical Analysis, Section 7.1.2

## **Model Checking & Diagnostics**

Refer to Appendix 11: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Adjusted means and the corresponding 95% confidence intervals will be presented by visit.
- The estimated adjusted means will be presented using the observed marginal distribution of the sample covariates (OM option in LSMEANS statement).
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used (DDMF=KR).
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line.
- Change from the baseline at each Visit X will be calculated by (Estimated Score at Visit X minus Estimated Score at Baseline) and the corresponding 95% confidence intervals.
   Adjusted means at each visit will also be presented.
- Plots of LS means change from baseline in SGRQ Score and 95% confidence intervals from the model will be generated by visit.

#### **On-treatment Phase**

See Primary Efficacy Statistical Analysis, Section 7.1.2

#### **Secondary Statistical Analyses**

#### Secondary Endpoint(s)

- Frequency of clinically significant asthma exacerbations over 32 week treatment
- Frequency of exacerbations requiring ED visit/hospitalization during the 32 week treatment period
- Frequency of exacerbations requiring hospitalization during the 32 week treatment period

#### Model Specification

- The frequency of clinically significant exacerbations will be analysed using Negative Binomial regression via generalised estimating equations with a covariate of time period (pre-, postmepolizumab).
- Exacerbations separated by less than 7 days will be treated as a continuation of the same exacerbation.
- The pre-mepolizumab exacerbation values (in the 12 months prior) will be obtained at screening, while the post-meplizumab exacerbation values will be observed during the study.
- The variance of the mean estimate will be corrected for within-subject correlation. The logarithm of time on treatment will be used as an offset variable.

#### **Model Checking & Diagnostics**

Refer to Appendix 11: Model Checking and Diagnostics for Statistical Analyses.

#### **Secondary Statistical Analyses**

#### **Model Results Presentation**

Adjusted exacerbation rate and the corresponding 95% confidence interval will be presented.

#### **On-treatment Phase**

- All subjects in the ITT population will be included within this analysis.
- All data collected up to and including Week 32 from patients, including those who have discontinued study treatment, will be included in the analysis.
- An On-Treatment "de jure" analysis will also be performed which does not consider any data collected following treatment discontinuation (see On-Treatment definition within Section 10.4).

## **Sensitivity and Supportive Statistical Analyses**

 The On-Treatment "de jure" analysis will be also performed with a subset of patients who were on omalizumab for more than 12 months.

# **Secondary Statistical Analyses**

## Secondary Endpoint(s)

• Ratio to baseline in blood eosinophil count at week 32

# **Model Specification**

- See Primary Efficacy Statistical Analysis, Section 7.1.2
- A log-transformation will be applied to blood eosinophil count data prior to analysis.
- If a blood eosinophil count of zero is reported, it will be imputed with half of the lowest possible blood eosinophil count, where applicable, prior to log transforming the data (Note: this imputation has typically been 0.5 \* 0.01 GI/L = 0.005 GI/L for previous mepolizumab studies).

#### **Model Checking & Diagnostics**

Refer to Appendix 11: Model Checking and Diagnostics for Statistical Analyses...

#### **Model Results Presentation**

- Adjusted means and the corresponding 95% confidence intervals will be presented by visit.
- Plots of LS means ratio to baseline in blood eosinophil count and 95% confidence intervals from the model will be generated by visit.

#### **On-treatment Phase**

- All subjects in the ITT population will be included within this analysis.
- All data collected up to and including Week 32 from patients, including those who have discontinued study treatment, will be included in the analysis.
- An On-Treatment "de jure" analysis will also be performed which does not consider any data collected following treatment discontinuation (see On-Treatment definition within Section 10.4.

#### Other Statistical Analyses

#### Other Endpoint

 Percentage of subjects achieving a 0.5-point or greater reduction from baseline in ACQ-5 score at Week 32

#### **Results Presentation**

- The number and percentage of subjects achieving a 0.5-point or greater reduction in ACQ-5 Score compared to baseline will be presented for each visit.
- The number of subjects with a missing ACQ-5 Score at each visit will be presented in a separate category.

#### **On-treatment Phase**

See Primary Efficacy Statistical Analysis, Section 7.1.2

## **Other Statistical Analyses**

#### Other Endpoint

 Percentage of subjects achieving a 4-point or greater reduction from baseline in SGRQ score at Week 32

#### **Results Presentation**

- The number and percentage of subjects achieving a 4-point or greater reduction in SGRQ Total score compared to baseline will be presented for each visit.
- The number of subjects with a missing SGRQ Total Score at each visit will be presented in a separate category.

#### **On-treatment Phase**

See Primary Efficacy Statistical Analysis, Section 7.1.2

## **Other Statistical Analyses**

## Other Endpoint

• Mean change from baseline in pre- and post- bronchodilator FEV1 at Week 32

#### **Model Specification**

See Primary Efficacy Statistical Analysis, Section 7.1.2

#### **Model Checking & Diagnostics**

• Refer to Appendix 11: Model Checking and Diagnostics for Statistical Analyses.

#### Model Results Presentation

- Adjusted means and the corresponding 95% confidence intervals will be presented by visit
- The estimated adjusted means will be presented using the observed marginal distributions of the sample covariates (OM option in LSMEANS statement).
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used (DDMF=KR).
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line.
- Change from the baseline at each Visit X will be calculated by (Estimated Score at Visit X minus Estimated Score at Baseline) and the corresponding 95% confidence intervals.
   Adjusted means at each visit will also be presented.
- Plots of Least Squares (LS) mean change from baseline pre- and post bronchodilator FEV1 and 95% confidence intervals from the model will be generated at each visit.

#### **On-treatment Phase**

See Primary Efficacy Statistical Analysis, Section 7.1.2

#### **Other Statistical Analyses**

#### Other Endpoint

- Subject rated response to therapy at Week 32
- Clinician rated response to therapy at Week 32

#### **Results Presentation**

- The number and percentage of subjects in each response category will be presented for each visit.
- The number of subjects with a missing responses at each visit will be presented in a separate category.

#### **On-treatment Phase**

 An On-Treatment "de jure" analysis will also be performed which does not consider any data collected following treatment discontinuation (see On-Treatment definition within Section 10.4).

#### Other Statistical Analyses

#### Other Endpoint

Mean change from baseline in Treatment Satisfaction Questionnaire for Medication (TSQM-9)

#### **Model Specification**

 The Mean Change at Week 32 will be tested to see if it is significantly different from zero using Wilcoxon signed-rank test

#### **Model Checking & Diagnostics**

 Check for the extreme outliers by plotting the differences between TSQM-9 at Week 32 and Baseline

#### **Model Results Presentation**

- Summary Statistics will be represented by study visit
- The mean change at Week 32 will presented with the corresponding 95% CI and p-value in the table
- The mean change at Week 32 will presented with the corresponding 95% CI in the figure

#### **On-treatment Phase**

 An On-Treatment "de jure" analysis will also be performed which does not consider any data collected following treatment discontinuation (see On-Treatment definition within Section 10.4)

#### **Other Statistical Analyses**

#### Other Endpoint

Change from baseline in inflammatory biomarkers expression at week 32.
 The following biomarker parameters will be reported:
 CCL13, CCL17, ECP, EDN, Eotaxin1, Total IL-5, IL-13, MDC, Periostin, TSLP

#### **Model Results Presentation**

- A log-transformation will be applied to each biomarker parameter prior to analysis.
- Summary Statistics will be represented by study visit, including ratio to baseline
- See Section 10.6.4 for further information regarding biomarker results below the lower limit of quantification

#### **On-treatment Phase**

 An On-Treatment "de jure" analysis will also be performed which does not consider any data collected following treatment discontinuation (see On-Treatment definition within Section 10.4).

# 8.2. Safety Analyses

# 8.2.1. Overview of Planned Analyses

The safety analyses will be based on the Intent-To-Treat (ITT) population, unless otherwise specified in Appendix 13: List of Data Displays. The safety displays to be created as part of the RAP include all the required and relevant displays identified as per the RAP Core Safety Reporting Template Version 1.0.

Table 6 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 13: List of Data Displays.

Adverse events will be coded using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA).

Table 6 Overview of Planned Adverse Event Analyses

| Endpoint / Parameter/ Display Type | | Absolute | |
|---|---|---|---|
| | Sun | nmary | Individual |
| | Т | F | L |
| Exposure | | _ | |
| Number of treatments administered and time on-treatment | Υ | | Υ |
| Adverse Events (AEs) | | | |
| Overview of Adverse Events | Υ | | |
| AEs by SOC and Maximum Intensity | Υ | | Υ |
| Common Adverse Events by Overall Frequency [1] | Υ | | |
| All Drug-Related AEs by SOC and Maximum Intensity | Υ | | |
| AEs on the Day of Dosing | Υ | | |
| AEs by the Age Group (<18 year, ≥18 years) | Υ | | |
| AEs by Highest Antidrug Antibody Result At Any Time Post Baseline | Υ | | |
| Number of subjects & occurrences of common <sup>[1]</sup> non-serious AEs by SOC and PT | Y | | |
| Subject Numbers for Individual AEs | | | Υ |
| Relationship between AE SOCs, PT & verbatim text | | | Υ |
| Serious and Other Significant AEs | | | |
| Fatal Serious AEs | Υ | | Υ |
| Non-Fatal Serious AEs | Υ | | Υ |
| Serious AEs by SOC | Υ | | |
| Reasons for Considering as a Serious AE | | | Υ |
| Drug-Related Serious AEs by SOC and Maximum Intensity | Υ | | |
| AEs Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment by Overall Frequency | Y | | Υ |
| Number of Subjects and Occurrences of Serious, Drug-Related Serious, Fatal Serious, and Drug-Related Fatal Serious AEs | Y | | |
| Adverse Events of Special Interest (AESI) (On-Treatment) [2] | | | |
| Anaphylaxis | Υ | | Υ |
| Systemic Allergic/Hypersensitivity and Non-allergic Reactions | Υ | | Υ |

| Endpoint / Parameter/ Display Type | | Absolute | |
|---|---|---|---|
| | Sur | nmary | Individual |
| | T | F | L |
| Systemic Allergic/Hypersensitivity Reactions | Υ | | |
| Systemic Non-allergic Reactions | Υ | | |
| Local Injection Site Reactions | Y | | Y |
| Opportunistic Infections | Y | | Υ |
| Malignancies | Y | | Y |
| Serious Cardiac, Vascular and Thromboembolic Events | Y | | Υ |
| Serious Ischemic Events | Y | | Υ |
| Cardiovascular Events | • | • | • |
| All Cardiovascular Events | Υ | | Υ |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Display generated, SOC=System Organ Class, PT=Preferred Term.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] Common AEs will be defined as AEs with frequency ≥3% (prior to rounding to nearest percent).
- [2] On-treatment Summary Profiles of each type of AE of Special Interest will also be presented.

#### 8.2.2. Adverse Events of Special Interest

Adverse events of special interest (AESIs) are adverse events associated with the identified and potential risks of mepolizumab. AESIs of anaphylaxis reactions, systemic reactions, and local injection site reactions are collected via targeted eCRF within the study. Events captured on the eCRF as systemic reactions will be further categorized as allergic/hypersensitivity reactions or non-allergic reactions. Events with preferred terms such as injection related reaction or administration related reaction will be considered non-allergic reactions. All remaining events will be considered allergic/hypersensitivity reactions.

AESIs of opportunistic infections, malignancies, serious CVT events and serious ischemic events will be identified from a list of relevant preferred terms maintained within a project level reference dataset created based on the MedDRA dictionary available at the time of database freeze for this study, further details of how relevant preferred terms are identified are given in the Program Safety Analysis Plan (PSAP).

Separate summary tables showing the number and percent of subjects with each type of AESI, broken down by preferred term will be created. Information will be reported as part of the standard AE tables for AESIs of infections, serious infections, neoplasms, cardiac disorders and serious cardiac disorders.

For each type of AESI a profile summary table will be produced containing information which would include, but not be limited to, the number of occurrences of the event, event characteristics, time to onset, intensity, outcome and action taken.

A listing of any subjects with systemic events identified by the investigators as meeting the criteria for anaphylaxis as outlined by the 2006 Joint National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network Second Symposium on

Anaphylaxis [Sampson, 2006] will be provided. Adverse events experienced on a day of dosing will be summarised and presented by SOC and preferred term.

A listing of all adverse events experienced by subjects who have had at least one investigator defined systemic reaction will be provided.

Cardiovascular events will be captured on targeted CV event pages of the CRF for the following AEs and SAEs:

- Myocardial infarction/unstable angina
- Congestive heart failure
- Arrhythmias
- Valvulopathy
- Pulmonary hypertension
- Cerebrovascular events/stroke and transient ischemic attack
- Peripheral arterial thromboembolism
- Deep venous thrombosis/pulmonary embolism
- Revascularization

## 8.2.3. Overview of Planned Clinical Laboratory Analyses

Safety analyses will be based on the Intent-To-Treat (ITT) population, unless otherwise specified in Appendix 13: List of Data Displays. The safety displays to be created as part of the RAP include all the required and relevant displays identified as per the RAP Core Safety Reporting Template Version 1.0.

Table 7 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 13: List of Data Displays.

Table 7 Overview of Planned Clinical Laboratory Analyses

| Endpoint / Parameter/ Display Type | | Abs | olute | Ch | Change from BL | |
|---|---|---|---|---|---|---|
| | Summary Individual | | | Summary | | Individual |
| | Т | F | L | T | F | L |
| Chemistry | | | | | | |
| Change from Baseline in Clinical Chemistry by Visit | | | | Υ | | |
| Chemistry Results (Change from Baseline Relative to Normal Range) | Υ | | | Υ | | |
| Hematology | | | | | | |
| Change From Baseline in Haematology by Visit | | | | Υ | | |
| Haematology Results (Change from Baseline Relative to Normal Range) | Υ | | | Υ | | |
| Hepatobiliary (Liver) | | | | | | |
| Liver Monitoring/Stopping Event Reporting | | | Υ | | | |
| Chemistry Results for Subjects Meeting Liver | | | Y | | | |

| Endpoint / Parameter/ Display Type | | Abs | olute | Ch | Change from BL | |
|---|---|---|---|---|---|---|
| | Summary Individual | | | Summary | | Individual |
| | Т | F | L | Т | F | L |
| Monitoring/Stopping Event Criteria | | | | | | |
| Medical Conditions for Subjects with Liver Stopping Events | | | Y | | | |
| Alcohol Intake for Subjects with Liver Stopping Events | | | Y | | | |
| Hepatobiliary Laboratory Abnormalities | Υ | | Y | | | |
| Scatter Plot of Maximum Post-Baseline vs. Baseline for ALT | | Υ | | | | |
| Scatter Plot of Maximum Post-Baseline ALT vs<br>Maximum Post-Baseline Total Bilirubin | | Υ | | | | |
| All Laboratory | | | | | | |
| All Laboratory Data for Subjects with any Value of Potential Clinical Concern | | | Y | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

# 8.2.4. Overview of Planned Other Safety Analyses

The safety analyses will be based on the Intent-To-Treat (ITT) population, unless otherwise specified in Appendix 13: List of Data Displays. The safety displays to be created as part of the RAP include all the required and relevant displays identified as per the RAP Core Safety Reporting Template Version 1.0.

Table 8 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 13: List of Data Displays.

Table 8 Overview of Planned Other Safety Analyses

| Endpoint / Parameter/ Display Type | | Abs | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| | Sum | Summary Individual | | Summary | | Individual |
| | Т | F | L | T | F | L |
| ECG | | | | | | |
| ECG Findings | Υ | | Υ | | | |
| Change from Baseline in ECG Values by Visit | | | | Υ | | |
| Actual and Change From Baseline QTc(F) Values by Category | Υ | | | Y | | |
| Actual and Change From Baseline QTc(B) Values by Category | Υ | | | Y | | |

| Endpoint / Parameter/ Display Type | | Abso | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| | Summary | | Individual | Summary | | Individual |
| | Т | T F L | | T | F | L |
| Vital Signs | | | | | | |
| Change from Baseline in Vital Signs by Visits | | | | Υ | | |
| Immunogenicity | | | | | | |
| Immunogenicity (ADA and NAb results) | Υ | | Υ | | | |
| Treatment Emergent ADA results | Υ | | | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

## 8.2.4.1. Immunogenicity

Immunogenicity is a measure of the immune response to a therapeutic drug (e.g. a monoclonal antibody) resulting in generation of anti-drug antibodies. Clinical samples are tested in a sequence of binding anti-drug antibody (ADA) and neutralising antibody assays:

- a) Screening assay. Each sample is tested for the presence of anti-drug antibodies (ADA assay) and initially declared positive or negative according to assay cut-off criteria. Negative samples are not tested further. Positive samples are then tested in the confirmation ADA assay.
- b) Confirmation assay. Each positive sample from the screening assay is either confirmed positive in this assay (ADA assay), or is declared negative and are not tested further. Positive ADA samples are then tested in the titer assay and neutralization (NAb) assay.
- c) Titration assay. Each positive sample from the ADA confirmation assay is serially diluted to provide a titre, corresponding to the highest dilution factor that still yields a positive test result.
- d) Neutralising assay. Each positive sample from the ADA confirmation assay is tested with the neutralising antibody assay and found as either positive or negative in this assay (NAb assay).

The mepolizumb ADA (screening/confirmation/titration) assay version 2011N122789 is performed at a Alliance Pharma (method 120711M01.V02). The mepolizumb Nab assay version 2011n129752 is being performed within GSK.

- A table will be produced summarising the number and percentage of negative and confirmed positive subjects ADA samples by treatment group and visit in the ITT population. The table will also summarise the highest assay result obtained postbaseline for each subject.
- A similar table will also be produced summarising results for the neutralising antibody assay in the ITT Population, by treatment group and visit.

- An additional summary of treatment emergent positive confirmatory binding antibody assay and results in the subset of subjects who did not have a positive confirmatory binding antibody assay result prior to the first dose of study treatment will also be presented.
- All immunogenicity results (i.e. ADA screening and confirmatory assay results, titre values, neutralising antibody results and observed mepolizumab concentration) will be listed.

## 9. REFERENCES

GlaxoSmithKline Document Number 2015N243304\_00 Study ID 204471. A multicentre, open label, single arm, 32-week treatment study in subjects with severe eosinophilic asthma not optimally controlled with current omalizumab treatment who are switched from omalizumab to mepolizumab 100mg subcutaneous (study number 204471-the OSMO study). Report Date 19-OCT-2015.

GlaxoSmithKline Document Number 2015N243304\_01 Study ID 204471. A multicentre, open label, single arm, 32-week treatment study in subjects with severe eosinophilic asthma not optimally controlled with current omalizumab treatment who are switched from omalizumab to mepolizumab 100mg subcutaneous (study number 204471-the OSMO study). Report Date 23-MAR-2016.

GlaxoSmithKline Document Number n/a Study ID Across Studies. Program Safety Analysis Plan for Mepolizumab (SB240563). Report Date 31-Mar-2017.

Juniper EF, O'Byrne PM, Guyatt GH, Ferrie PJ, King DR. Development and validation of a questionnaire to measure asthma control. *Eur Respir J.* 1999;14:902–907.

Juniper EF, Svensson K, Mork AC, Stahl E. Measurement properties and interpretation of three shortened versions of the asthma control questionnaire. *Respiratory Medicine*. 2005;99:553–558.

Quanjer P., Stanojevic S., Cole T., Baur X., Hall G., Culver B., Enright P., Hankinson J., Ip M., Zheng J., Stocks J., & ERS Global Lung Function Initiative. Multi-ethnic reference values for spirometry for the 3-95-yr age range: The global lung function 2012 equations. *European Respiratory Journal*. 2012;40(6):1324-1343.

Quanjer P., Stanojevic S., Cole T., Baur X., Hall G., Culver B., Enright P., Hankinson J., Ip M., Zheng J., Stocks J., & ERS Global Lung Function Initiative. Multi-ethnic reference values for spirometry for the 3-95-yr age range: The global lung function 2012 equations - Supplemental Material. *European Respiratory Journal*. 2012;40(6):1324-1343.

Sampson HA, Munoz-Furlong A, Campbell RL et al. Second Symposium on the definition and management of anaphylaxis: Summary Report.Second National Institute of Allergy and Infectious Disease / Food Allergy and Anaphylaxis Network Symposium. *Journal of Allergy and Clinical Immunology*. 2006;117:391-397.

Winthrop KL, Novosad SA, Baddley JW, et al. Opportunistic infections and biologic therapies in immune-mediated inflammatory diseases - consensus recommendations for infection reporting during clinical trials and postmarketing surveillance. *Ann Rheum Dis*. 2015;0:1–10.

Atkinson MJ, Kumar R, Cappelleri JC, Hass SL. Hierarchical construct validity of the treatment satisfaction questionnaire for medication (TSQM version II) among outpatient pharmacy consumers. *Value Health.* 2005;8(Suppl 1):S9-S24.

# 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4 | : Analysis Populations |
| Section 10.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.2 | Appendix 2: Time & Events |
| Section 10.3 | Appendix 3: Assessment Windows & Visit Slotting |
| Section 10.4 | Appendix 4: Treatment Phases |
| Section 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| | Study Treatment & Subgroup Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.6 | Appendix 6: Derived and Transformed Data |
| | General |
| | Study Population |
| | Efficacy |
| | Safety |
| Section 10.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 10.8 | Appendix 8: Values of Potential Clinical Importance |
| | Laboratory Values |
| Section 10.9 | Appendix 9: Multicenter Studies |
| Section 10.10 | Appendix 10: Examination of Covariates and Subgroups |
| Section 10.11 | Appendix 11: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP App | |
| Section 10.12 | Appendix 12: Abbreviations & Trade Marks |
| Section 10.13 | Appendix 13: List of Data Displays |
| Section 10.14 | Appendix 14: Example Mock Shells for Data Displays |

# 10.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

# 10.1.1. Exclusions from Per Protocol Population

Subjects with protocol deviations considered to potentially have an effect on efficacy will be excluded from the Per Protocol (PP) population. Determination of the Per Protocol population will be performed before the database is frozen. The reason for the exclusion of any subject will be documented.

A subject meeting any of the following criteria will be excluded from the Per Protocol population:

| Number | Exclusion Description |
|---|---|
| 01 | Inclusion criteria # 2 – Insufficient evidence of asthma for ≥2 years that meets the National Heart and Lung Institute guidelines or GINA guidelines |
| 02 | Inclusion criteria # 3 – No persistent airflow obstruction as indicated by For subjects ≥18 years of age at Visit 1, a pre-bronchodilator FEV1 <80% predicted [Quanjer, 2012] recorded at Visit 1. For subjects 12-17 years of age at Visit 1, a pre-bronchodilator FEV1 <90% predicted [Quanjer, 2012] OR FEV1/FVC ratio <0.8 recorded at Visit 1. |
| | Inclusion criteria # 4 – No eosinophilic airway inflammation as defined by: |
| 03 | <ul> <li>Peripheral blood eosinophil level of ≥300 cells/µL that is related to asthma<br/>demonstrated in the 12 months prior to visit 1 OR</li> </ul> |
| | <ul> <li>Peripheral blood eosinophil level of ≥150 cells/µL demonstrated at Visit 1 that is<br/>related to asthma</li> </ul> |
| 04 | Inclusion criteria # 5 – Absence of evidence of a well-documented requirement for regular treatment with high dose ICS (equivalent to ≥880µg/day fluticasone propionate (FP) (exactuator) or equivalent daily in adults and ≥440µg/day FP (ex-actuator) or equivalent daily for subjects aged 12-17) in the 12 months prior to Visit 1 [Note: For ICS/LABA combination preparations, the highest approved maintenance dose in the local country will meet this ICS criterion.] |
| 05 | Inclusion criteria # 6 – Absence of current treatment with an additional controller medication, besides ICS, for at least 3 months or a documented failure in the past 12 months of an additional controller medication for at least 3 successive months [e.g., long-acting beta-2-agonist (LABA), leukotriene receptor antagonist (LTRA), or theophylline] |
| 06 | Inclusion criteria # 7 – Asthma symptoms not uncontrolled at Visit 1, as defined by an ACQ-5 score of <1.5. |
| 07 | Inclusion criteria # 8 – Not receiving Omalizumab treatment based on weight and IgE levels, for at least the 4 months prior to Visit 1. |
| 08 | Inclusion criteria # 9 – No history of two or more exacerbations requiring treatment with systemic corticosteroids (intramuscular, intravenous, or oral) in the 12 months prior to Visit 1 despite the use of high-dose ICS. [Note: For subjects receiving omalizumab for ≥8 months, at least one exacerbation must have occurred while on omalizumab treatment. For subjects receiving maintenance oral corticosteroids, the corticosteroid treatment for the exacerbations must have been a two-fold dose increase or greater.] |
| 09 | Continuation to treatment criteria # 1 – Asthma symptoms not uncontrolled at Visit 2, as |

| Number | Exclusion Description |
|---|---|
| | defined by an ACQ-5 score of <1.5. |
| 10 | Continuation to treatment criteria # 2 – Subjects who experience an asthma exacerbation during run-in who have not returned to their baseline asthma status within one week of Visit 2. |
| 11 | Continuation to treatment criteria # 3 – Any subject with changes in the dose or regimen of ICS, and/or additional controller medication (except for treatment of an exacerbation) during the run-in period. |
| | Continuation to treatment criteria # 4 – Subjects who do not receive their last dose of Omalizumab during the correct period, as defined by: |
| 12 | <ul> <li>For subjects receiving omalizumab every 4 weeks, their last dose is received &lt;3<br/>or &gt;5 weeks prior to Visit 2.</li> </ul> |
| | <ul> <li>For subjects receiving omalizumab every 2 weeks, their last dose is received &lt;1<br/>or &gt;3 weeks prior to Visit 2.</li> </ul> |
| 13 | Any subject with changes in the dose or regimen of baseline ICS, and/or additional controller medication during open-label treatment. |
| | N.B. This excludes the use of OCS for the treatment of an asthma exacerbation. |
| 14 | Use of any prohibited medication during the study [1]. |
| 15 | Receiving the incorrect study treatment at any point during the study. |

#### NOTES

• [1] See Protocol Section 6.8.2 for the list of prohibited medications within this study.

2017N328770\_00 **CONFIDENTIAL** 204471

# 10.2. Appendix 2: Time & Events

# 10.2.1. Protocol Defined Time & Events

Table 9 Time and Events Table

| Procedures | Pre-<br>screen <sup>1</sup> | Screen<br>Run-in | | | | | | | | | Exit Visit/<br>Early withdrawal<br>Visit³ |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| Week | -6 to -4 | -4 to -1 | 0 | 4 | 8 | 12 | 16 | 20 | 24 | 28 | 4 weeks post last dose ±7 days |
| Informed Consent <sup>2</sup> | Х | | | | | | | | | | |
| Subject Demography | х | | | | | | | | | | |
| Medical History | | Х | | | | | | | | | |
| Asthma History (including triggers) | х | X | | | | | | | | | |
| Therapy History <sup>4</sup> | | Х | | | | | | | | | |
| Smoking History | | Х | | | | | | | | | |
| Cardiovascular History/Risk<br>Factors | | X | | | | | | | | | |
| Inclusion/Exclusion Criteria | | Х | | | | | | | | | |
| Continuation to treatment Criteria | | | х | | | | | | | | |
| Efficacy Assessments <sup>5</sup> | | | | | | | | | | | |
| ACQ-5 | | X | Х | Х | Х | Х | Х | Х | Х | Х | х |
| Exacerbation review | Х | Х | Х | Х | х | Х | Х | Х | Х | Х | Х |
| Spirometry including pre- and post bronchodilator FEV <sub>1</sub> , FVC <sup>6</sup> | | Х | X | | | х | | | х | | х |
| Health Outcome | | | | | | | | | | | |
| Assessments <sup>5</sup> | | | | | | | | | | | |
| SGRQ | | | X | | | X | | | Х | | X |

| Procedures | Pre-<br>screen <sup>1</sup> | Screen<br>Run-in | | Exit Visit/<br>Early withdrawal<br>Visit <sup>3</sup> | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| Week | -6 to -4 | -4 to -1 | 0 | 4 | 8 | 12 | 16 | 20 | 24 | 28 | 4 weeks post last dose ±7 days |
| Clinician & Subject rated response to therapy | | | | | х | | х | | х | | х |
| Treatment Satisfaction with Medication Questionnaire (TSQM-9) | | Х | | | | | | | | | х |
| Exit Interview <sup>7</sup> | | | | | | | | | | | X |
| Safety Assessments <sup>5</sup> | | | | | | | | | | | |
| Concomitant Medication | X | X | X | x | X | X | X | X | x | X | X |
| Physical Examination, including nasal exam | | X | | | | | | | | | x |
| Vital Signs | | X | X | X | X | X | X | X | X | X | X |
| 12 lead ECG | | X | | | | X | | | | | х |
| Adverse Events | | X | X | X | X | X | X | X | X | X | X |
| Serious Adverse Events | х | X | X | X | X | X | X | X | X | X | X |
| Laboratory Assessments <sup>5</sup> | | | | | | | | | | | |
| Haematology with differential | | х | X | X | X | X | Х | X | X | X | X |
| Clinical Chemistry (incl. LFT) | | X | X | X | X | X | | | X | | X |
| Parasitic Screening <sup>8</sup> | | X | | | | | | | | | |
| Pharmacogenetic sample9 | | | | χ , | | | | | | | |
| Pregnancy test <sup>10</sup> | | U | U | U | U | U | U | U | U | U | U |
| HBsAg and hepatitis C antibody <sup>11</sup> | | Х | | | | | | | | | |
| Immunogenicity sample | | | х | | | х | | | | х | х |
| Biomarker sample | | Х | х | | х | | | | | | x |

| Procedures | Pre-<br>screen <sup>1</sup> | Screen<br>Run-in | Treatment (visit window is ±7days) | | | | | | | | Exit Visit/<br>Early withdrawal<br>Visit³ |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| Week | -6 to -4 | -4 to -1 | 0 | 4 | 8 | 12 | 16 | 20 | 24 | 28 | 4 weeks post last dose ±7 days |
| Investigational product (Mepolizumab) and rescue medication | | | , | | | | | | | | |
| Administer mepolizumab. Contact RAMOS NG to register dispensing visit. | | | х | х | х | х | х | х | х | х | |
| Albuterol/salbutamol dispensed (as needed) | | X | х | х | х | х | Х | Х | х | х | |
| Collect dispensed albuterol/salbutamol | | | х | Х | х | х | Х | Х | х | х | х |
| eCRF/<br>paper diary/worksheet | | | | | | | | | | | |
| Complete eCRF | х | х | Х | Х | Х | Х | Х | Х | Х | Х | X |
| Dispense paper diary/worksheet | Х | Х | х | Х | х | х | Х | Х | х | х | |
| Collect/review paper diary/worksheet | | X | х | X | Х | х | Х | X | х | х | X |

- 1. Pre-screen Visit 0 must be completed prior to Visit 1 (Screening). It can be completed on the same day as Visit 1 or at up to 2 weeks prior to Visit 1.
- 2. Subjects will be assigned a subject number at the time ICF signed. The ICF must be signed before any study procedures including medication wash out period(s).
- 3. Exit Visit may be completed 3 to 5 weeks post last dose.
- 4. Therapy history to include a detailed review of prior biologics received for treatment of asthma, including omalizumab dose and regimen and prior investigational therapies e.g anti-IL5 or anti-IL13 preparations.
- 5. All study efficacy, safety and all patient reported questionnaires must be completed prior any study procedure.
- 6. Spirometry to include pre- and post bronchodilator FEV1 from V2.
- 7. Exit interview will be conducted only in a subset of sites and in a subset of subjects who choose to participate in the Exit interview. Subjects must be consented prior to interview
- 8. Parasitic screening is only required in countries with high-risk or for subjects who have visited high-risk countries in the past 6 months. Sites should use local laboratories.
- 9. Pharmacogenetic sample may be drawn at Visit 2 or any at any visit after.
- 10. Pregnancy test, U= urine
- 11. Hepatitis B Surface Antigen and Hepatitis C antibody. (if hepatitis C antibody is positive, hepatitis C will be confirmed by PCR)
## 10.3. Appendix 3: Assessment Windows & Visit Slotting

#### 10.3.1. Assessment Windows

Clinic visits are scheduled to take place as specified in Appendix 2: Time & Events. Measurements outside visit windows will not be excluded from analyses. For all clinic visits, nominal visit days and times will be used for reporting, such that if a subject recorded values that were outside of the  $\pm 7$  day window for a visit they will still be reported under that visit.

## 10.3.2. Early Withdrawal / Treatment Discontinuation Visits

If a subject withdraws from the study at a scheduled visit (i.e. completes an Early Withdrawal or Treatment Discontinuation Visit), where endpoint data were scheduled to be collected, the data will be summarised and analysed (as appropriate) together with data from subjects who did not withdraw from the study. If a subject withdraws from the study at a scheduled visit at which endpoint data were not scheduled to be collected, or if a subject withdraws between scheduled visits, data will be slotted to the nearest adjacent visit where the endpoint data was scheduled to be collected (if data at that visit were not recorded) according to the Time and Events schedule (Appendix 2: Time & Events).

For example, if a subject prematurely withdraws from the study and completed the Early Withdrawal Visit at Visit 6 (Week 16) and completes an Early Withdrawal Visit which includes an  $FEV_1$  assessment, the  $FEV_1$  data collected will need to be re-assigned to an adjacent visit where  $FEV_1$  data is scheduled for collection. In this case the  $FEV_1$  data will be reassigned to Visit 5 (Week 12) (if data at that visit were not recorded) as this is the closest nominal visit at which collection of  $FEV_1$  data is scheduled.

#### 10.3.3. Unscheduled Visits

For unscheduled visits, similar logic will be applied. If a subject has an unscheduled assessment then this data would be slotted to the closest adjacent scheduled visit but only if information already exists at that visit. If an unscheduled visit occurred between two scheduled visits for which data has been reported, then the data from the unscheduled visit will remain in the unscheduled visit and will not be used in summary tables and analyses (except for endpoints using any post-baseline data) but will be presented in any relevant listings.

## 10.4. Appendix 4: Treatment Phases

## 10.4.1. Treatment Phases (Exacerbations)

Exacerbation data will be classified according to time of occurrence/assessment relative to the first and last date of mepolizumab and the attendance dates of specific visits.

| Treatment Phase | Definition |
|---|---|
| Pre-Treatment | Date & time < First dose of mepolizumab |
| On-Treatment | Subjects completing treatment and completing the study: |
| | First dose of mepolizumab ≤ Date & time ≤ Visit 10 (Exit Visit)* visit date |
| | Subjects discontinuing study treatment/withdrawing early from the study: |
| | First dose of mepolizumab ≤ Date & time ≤ Earliest of (1) Last dose of mepolizumab + |
| | 28 days or (2) Early Withdrawal/Treatment Discontinuation visit date |
| Off-Treatment | Subjects completing treatment and completing the study: |
| | Date & time > Visit 10 (Exit Visit)* visit date |
| | Subjects discontinuing study treatment/withdrawing early from the study: |
| | Date & time > Earliest of : |
| | (1) Last dose of mepolizumab + 28 days or |
| | (2) Early Withdrawal/Treatment Discontinuation visit date |

<sup>\*</sup> Data may be considered off treatment if beyond acceptable protocol defined limits.

## 10.4.2. Treatment Phases (Visit Based Efficacy Data)

Efficacy data collected at scheduled visits (including: Questionnaires, PFT, Blood Eosinophils and Biomarkers) will be classified according to time of occurrence/assessment relative to the first and last date of mepolizumab and the attendance dates of specific visits.

| Treatment Phase | Definition |
|---|---|
| Pre-Treatment | Visit date/time ≤ First dose of mepolizumab |
| On-Treatment | Subjects completing treatment and completing the study: |
| | Visit date/time < First dose of mepolizumab ≤ Visit 10 (Exit Visit)* visit date/time |
| | Subjects discontinuing study treatment/withdrawing early from the study: |
| | Visit date/time < First dose of mepolizumab ≤ Earliest of (1) Last dose of mepolizumab |
| | + 28 days or (2) Early Withdrawal/Treatment Discontinuation visit date date/time |
| Off-Treatment | Subjects completing treatment and completing the study: |
| | Date & time > Visit 10 (Exit Visit)* visit date/time |
| | Subjects discontinuing study treatment/withdrawing early from the study: |
| | Date & time > Earliest of: |
| | (1) Last dose of mepolizumab + 28 days or |
| | (2) Early Withdrawal/Treatment Discontinuation visit date/time |

<sup>\*</sup> Data may be considered off treatment if beyond acceptable protocol defined limits.

## 10.4.3. Treatment Phases (Adverse Events)

Adverse events will be classified according to time of occurrence relative to the first and last date of the study treatment.

| Treatment Phase | ment Phase Definition | | |
|---|---|---|---|
| Pre-Treatment | AE Onset Date & time < First dose of mepolizumab | | |
| | If mepolizumab treatment is never started then all AEs will be classified as pre- | | |
| | treatment. | | |
| On- Treatment | - Treatment First dose of mepolizumab ≤ AE Onset Date & time ≤ Last dose of mepolizumab + | | |
| days If an AE start date is missing or partial then the AE will be considered on-treatn unless there is evidence to the contrary (e.g. month/year of onset date is prese | | | |
| | | | earlier than the month/year of First dose of mepolizumab). |
| | | Post-treatment | AE Onset Date & time > Last dose of mepolizumab + 28 days |

#### 10.4.3.1. Adverse Event Data Derivations

| Treatment State | Definition |
|---|---|
| Onset Time<br>Since 1st Dose<br>(Days) | If Treatment Start Date > AE Onset Date = AE Onset Date - First dose of mepolizumab If Treatment Start Date ≤ AE Onset Date = AE Onset Date - First dose of mepolizumab +1 |
| | If Treatment Start Date or AE Onset Date is missing = missing. |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related If relationship is marked 'YES' on Inform/eCRF OR value is missing. | |

## 10.4.4. Treatment Phases (Concomitant Medications)

Concomitant medications will be classified according to time of occurrence relative to the first and last date of the study treatment.

| Treatment/Study Phase | Definition |
|---|---|
| Taken Before the Run-in | If Con-med Start Date < Date of Visit 1 |
| Taken During the Run-in | <ul> <li>If Con-med Start Date &lt; Date of Visit 1 and Con-med Stop Date ≤ Date of Visit 1, or</li> <li>If Date of Visit 1 ≤ Con-med Start Date &lt; First dose of mepolizumab</li> </ul> |
| Taken During<br>Treatment | <ul> <li>If Con-med Start Date &lt; First dose of mepolizumab and Con-med Stop Date ≥ First dose of mepolizumab or</li> <li>If First dose of mepolizumab≤ Con-med Start Date ≤ Last dose of mepolizumab+ 28 days</li> <li>If the con-med start or stop date is missing or partial then the con-med will be considered on-treatment unless there is evidence to the contrary (e.g. month/year of con-med stop date is present and is before the month/year of the first dose of mepolizumab).</li> </ul> |
| Started During<br>Treatment | Subset of con-meds Taken During Treatment for which: First dose of mepolizumab ≤ Con-med Start Date ≤ Last dose of mepolizumab + 28 days |
| Taken Post Treatment • Last dose of mepolizumab + 28 days < Con-med Stop Date | |

A medication will be summarised in every treatment/study phase in which it was taken,

so for example a medication that was started in the run-in and stopped during treatment will appear in both the during the run-in and during treatment tables.

# 10.5. Appendix 5: Data Display Standards & Handling Conventions

#### 10.5.1. Study Treatment & Subgroup Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| RandAll NG | | Data Displays for Reporti | ng |
| Code | Description | Description | Order [1] |
| 1 | Mepolizumab 100mg SC | Mepolizumab 100mg SC | 1 |

#### NOTES:

1. Order represents treatments being presented in TFL, as appropriate.

#### 10.5.2. Baseline Definition & Derivations

#### 10.5.2.1. Baseline Definition

- Baseline will be defined for all subjects who are within the ITT population.
- For all endpoints the baseline values for each assessment will be the latest available assessment prior to first dose of mepolizumab.
- Measurements on the same date as the first administration of mepolizumab will be considered
  within the baseline derivation if measurement time is not captured. Where the measurement
  time is captured this should be compared against the time of first receiving mepolizumab.

#### 10.5.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|----------------------|--------------------------|
| Change from Baseline | = Visit Value – Baseline |
| Ratio to Baseline | = Visit Value / Baseline |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.5.2.1 Baseline Definitions will be used for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.

#### 10.5.3. Reporting Process & Standards

| Reporting Process | |
|---|---|
| Software | |
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : uk1salx00175 |
| HARP Area | : /arenv/arprod/sb240563/mid204471/final01 |
| Quality Control (QC) Spread sheet | : /arenv/arprod/sb240563/mid204471/final01/documents |

#### **Reporting Process**

### **Analysis Datasets**

- Analysis datasets will be created according to CDISC standards.
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### **Generation of RTF Files**

RTF files will be generated only for summary tables.

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- The reported precision (decimal places) will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of decimal places.

#### Planned and Actual Time

- Reporting for tables, figures and formal statistical analyses :
  - Nominal visits (planned time relative to dosing) will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Scheduled visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings, summaries and statistical analyses.

#### **Unscheduled Visits**

When possible unscheduled assessments will be slotted to the closest adjacent scheduled visit. If an unscheduled visit occurs between two completed scheduled visits, the data from the unscheduled visit will not be used in summary tables which are based on by-visit assessments. The information from the unscheduled visit will be included in 'any time post-baseline' summaries and will also be presented in any relevant listings. See Section 10.3 for further details.

| Descriptive Summary Statistics | |
|--------------------------------|-------------------|
| Continuous Data | Defer to IDCL Sta |

| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
|---|---|
| Categorical Data | N (number of subjects in the treatment group), n (number of subjects with |

| Reporting Standards | |
|---|---|
| | non-missing values), frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

## 10.6. Appendix 6: Derived and Transformed Data

#### 10.6.1. General

## **Multiple Measurements at One Time Point**

- There are no scheduled multiple measurements, however, if multiple measurements are recorded at a given time point the following process will be followed, unless a process for selection of the measurement for the visit is specified:
- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables.

#### Study Day

- Calculated as the number of days from date of first dose of mepolizumab:
  - Ref Date = Missing
     Study Day = Missing
  - Ref Date < Date of first dose of mepolizumab</li>
     → Study Day = Ref Date Date of first dose of mepolizumab
  - Ref Data ≥ Date of first dose of mepolizumab →
     Study Day = Ref Date (Date of first dose of mepolizumab) + 1

## 10.6.2. Study Population

#### **Demographics**

#### Age

- Only year of birth was collected for subjects; actual birth data was not collected.
- GSK standard IDSL algorithms will be used for calculating age where the birth date of all subjects will be imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Each subject's derived age will be calculated as an integer value based on their imputed date of birth relative to the date of the subject's screening visit (Visit 1).
   [(30th June of the year of birth reported on eCRF – date of Screening)/365.25]

#### **Body Mass Index (BMI)**

• Calculated as Weight (kg) / Height (m)<sup>2</sup>

#### **Percent Predicted FEV1**

 FEV1 % of predicted normal will be derived using the Global Lung Function Initiative 2012 lookup tables which are based on the Quanjer equations [Quanjer, 2012] according to the Race/Ethnicity designations specified below:

| Collected Race <sup>[1]</sup> | Quanjer Designation |
|---|---|
| African American/African Heritage | African-American calculation will be applied |
| American Indian or Alaskan Native | Other calculation will be applied |

| Demographics | |
|---|---|
| Asian-Central/South Asian Heritage | South East Asian calculation will be applied |
| Asian-East Asian Heritage | North East Asian calculation will be applied |
| Asian-Japanese Heritage | Other calculation will be applied |
| Asian- Southeast Heritage | South East Asian calculation will be applied |
| Native Hawaiian or Other Pacific Islander | Other calculation will be applied |
| White-Arabic/North African Heritage | Caucasian calculation will be applied |
| White-White/Caucasian/European Heritage | Caucasian calculation will be applied |
| NOTES: | |
| <ol> <li>If multiple races are selected for a single sub</li> </ol> | ject then the "Other" calculation will be applied. |

#### FEV<sub>1</sub>/FVC Ratio

Pre- and post-bronchodilator FEV<sub>1</sub>/FVC ratio will be calculated as the ratio of the FEV<sub>1</sub> and FVC values.

#### Length of Omalizumab (Xolair) Use

Number of days exposed to Omalizumab (Xolair) will be calculated based on the formula:
 For subjects receiving Omalizumab (Xolair) monthly:

Duration of Exposure in Days = Last Omalizumab dose – (First Omalizumab dose) + 29 For subjects receiving Omalizumab (Xolair) twice monthly:

Duration of Exposure in Days = Last Omalizumab dose – (First Omalizumab dose) + 15

#### Baseline OCS daily dose

- Only corticosteroids administered via oral, intravenous (IV) and intramuscular (IM) routes are to be considered when calculating a subject's total daily prednisone/prednisolone asthma maintenance dose at baseline. All steroids administered via a sublingual route will also be considered as oral.
- The corticosteroid conversion factors shown below will be used, regardless of the route of administration, to scale each corticosteroid dose to a prednisone equivalent dose. These three routes of administration (oral, IV and IM) are to be considered equivalent as it has been noted that the bioavailability of methylprednisolone is considered to be roughly equivalent following administration as an oral, IV or IM steroid.

| Standardised Medication Name | Scaling Factor |
|---------------------------------|----------------|
| Betamethasone | 8.33 |
| Betamethasone Dipropionate | 8.33 |
| Betamethasone Sodium Phosphate | 8.33 |
| Cortisone | 0.2 |
| Cortisone Acetate | 0.2 |
| Cortivazol | 17 |
| Deflazacort | 0.833 |
| Dexamethasone | 6.67 |
| Dexamethasone Sodium Phosphate | 6.67 |
| Fludrocortisone Acetate | 0 |
| Hydrocortisone | 0.25 |
| Hydrocortisone Sodium Succinate | 0.25 |

| Demographics | |
|-------------------------------------|------|
| Hydrocortisone Sodium Phosphate | 0.25 |
| Meprednisone | 1 |
| Methylprednisolone | 1.25 |
| Methylprednisolone Acetate | 1.25 |
| Methylprednisolone Sodium Succinate | 1.25 |
| Methylprednisone | 1.25 |
| Methylprednisone Acetate | 1.25 |
| Methylprednisolone Sodium Succinate | 1.25 |
| Methylprednisone | 1.25 |
| Methylprednisone Acetate | 1.25 |
| Prednisolone | 1 |
| Prednisolone Acetate | 1 |
| Prednisolone Hemisuccinate | 1 |
| Prednisolone Sodium Succinate | 1 |
| Prednisone | 1 |
| Prednisone Acetate | 1 |
| Triamcinolone | 1.25 |
| Triamcinolone Acetonide | 1.25 |

## 10.6.3. Efficacy

#### **Patient Reported Outcomes/Questionnaires**

#### ACQ-5

- Each question on the ACQ-5 is scored on a 7-point scale from 0 = no impairment to 6 = maximum impairment. The questions are equally weighted and the ACQ-5 score will be the mean of the 5 questions, thus giving a score between 0 (totally controlled) and 6 (severely uncontrolled) [Juniper, 1999; Juniper, 2005].
- If a subject does not complete 1 of the 5 questions at a visit, then the ACQ-5 score will be the mean of the responses to the remaining 4 questions at that visit.
- If a subject does not complete more than 1 of the 5 questions at a visit, then their ACQ-5 score will be set to missing at that visit.
- A subject will be deemed a responder if the subject has a ≥0.5 reduction in ACQ score from Baseline. ACQ-5 Responder/Non-responder category will be missing if the overall ACQ-5 score is missing.

## St George's Respiratory Questionnaire (SGRQ)

- The SGRQ comprises 50 questions with a recall period of 4 weeks.
- Scores are expressed as the percentage of overall impairment with 100 equal to the worst possible health and 0 the best.
- Scoring of each domain of the SGRQ (Symptoms, Activity, Impacts) and the Total score are described in the St George's Respiratory Questionnaire Manual (Version 2.3).

#### **Patient Reported Outcomes/Questionnaires**

#### Treatment Satisfaction with Medication Questionnaire (TSQM-9)

- TSQM Scale scores range from 0 to 100, with higher scores indicating higher satisfaction. No computed score should be lower or higher than these limits. [Atkinson, 2005]
- Effectiveness scale: ([(ltem 1 + ltem 2 + ltem 3) 3] divided by 18) × 100
   If one item is missing: ([(Sum of ltem 1 + ltem 2 + ltem 3)) 2] divided by (12) × 100
- Convenience scale: ([Sum of Item 4 to Item 6) − 3] divided by 18) × 100 If one item is missing: ([(Sum of Item 4 to Item 6)) − 2] divided by (12) × 100
- Overall Satisfaction scale: First recode Item 9 = (Item 9 1) x 5/6
- Then: ([Sum of Item 7 to Item 9) 3] divided by (12) × 100
   If any one Item is missing: ([Sum of Item 7 to Item 9) 2] divided by (8) x 100

#### **Exacerbations**

An exacerbation of asthma as defined as:

Worsening of asthma which requires use of systemic corticosteroids<sup>1</sup> and/or hospitalisation and/or Emergency Department (ED) visits.

- 1For all subjects, i.v. or oral steroid (e.g., prednisone) for at least 3 days or a single IM CS dose is required. For subjects on maintenance systemic corticosteroids, at least double the existing maintenance dose for at least 3 days is required.
- Within each subject, exacerbations that occurred less than seven days apart will be collapsed
  into a single exacerbation. Exacerbations for which the collapsing has already been performed
  will be included in the summaries and analyses. Exacerbations will be displayed in listings as
  captured within the eCRF. Exacerbations which are collapsed into a single exacerbation will be
  highlighted.
- The collapsed exacerbation records will be constructed as follows:
  - Start date (ASTDT) is the start date of the first exacerbation in the series
  - End date (AENDT) is the end date of the last exacerbation in the series
  - Outcome (CEOUT) is the worst outcome in the series (worst to best is Fatal, Not Resolved, Resolved)
  - o Cause (EBCAUSE) is the cause associated with the first exacerbation in the series
  - Withdrawal due to exacerbation (EBWD), OCS taken for exacerbation (OCSEXB), corticosteroids taken for exacerbation (CTSEXB), hospitalization due to exacerbation (HSPEXB), emergency visit due to exacerbation (EREXB), and intubation for exacerbation (INTUBEXB) are set to 'Y' if any value for the respective variable in the series equals 'Y'
  - Number of telephone calls (TPCNUM), home day visits (HMDYVSN), home night visits (HMNTVSN), home day+night visits (HMDYNTV), office visits (OFCVSN), urgent care/outpatient visits (UCOUTVSN), emergency room visits (ERVSN), days in intensive care (ICSDYNUM), days in general ward (GWDYNUM) and days hospitalized (HSPDYNUM) are the sum of all of the values in the series for each respective variable

#### **Blood Eosinophils**

 Blood eosinophils will be log-transformed prior to analysis. Summary statistics will include geometric mean, and a measure of spread (SD or SE) on the natural log scale. • If a blood eosinophil count of zero is reported, it will be imputed with half of the lowest possible blood eosinophil count, where applicable, prior to log transforming the data (Note: this imputation has typically been 0.5 \* 0.01 GI/L = 0.005 GI/L for previous mepolizumab studies).

## 10.6.4. Safety

#### **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula:

  Duration of Exposure in Days = Last mepolizumab dose (First mepolizumab dose) + 29
- The extent of exposure will also be summarised as the number of study treatments administered

#### **Adverse Events**

#### **Adverse Events of Special Interest**

Section 8.2.2 provides a full list of AEs of special interest for this compound.

Adverse events of special interest (AESIs) of anaphylaxis reactions, systemic reactions, and local injection site reactions are collected via targeted eCRF. Systemic reactions with preferred terms such as injection related reaction or administration related reaction will be considered non-allergic reactions; those with other preferred terms will be considered allergic/hypersensitivity reactions. The AESIs of opportunistic infections, malignancies, serious CVT events and serious ischemic events will be identified from a list of relevant preferred terms maintained within a project level reference dataset; created based on the latest version of the MedDRA dictionary available at the time of database freeze for this study (See Program Safety Analysis Plan for additional details).

#### **ECG Parameters**

#### RR Interval

All ECG parameters required in this study will be databased, and therefore, further derivations will not be performed by Stats and Programming. The definitions of these parameters are given in this section.

- If RR interval (msec) is not databased, then RR can be derived as:
  - [1] If QTcB is machine read & QTcF is not provided, then :

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

If ECGs are manually read, the RR value should be a collected value and will not be derived.

#### **Corrected QT Intervals**

- When not databased, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- If RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as :

#### **ECG Parameters**

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}} \qquad QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

- Individual maximum QTc(F) and QTc(B) values will also be summarised by treatment group for each scheduled study visit to show the number of subjects with maximum values (msec) in the following categories:
  - <= 450</p>
  - 450 < to <= 480
  - 480 < to <= 500
  - > 500
- Additionally, individual maximum changes from baseline in QTc(F) and QTc(B) values will be summarised by treatment group for each scheduled study visit to show the number of subjects with maximum changes (msec) in the following categories:
  - < -60
  - $\geq$  -60 to < -30
  - $\geq$  -30 to < 0
  - $\geq$  0 to < 30
  - $\geq$  30 to < 60
  - ≥ 60

## **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database (values below the lower limit of quantification), where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the lower limit of quantification for that particular parameter will be used to impute the corresponding numeric value as half the lower limit of quantification for that measure (LLQ/2).
- The above imputation of half the lower limit of quantification for that measure (LLQ/2) will also be applied to all biomarker parameters.
- Regarding blood eosinophil laboratory data please reference Section 10.6.3.

# 10.7. Appendix 7: Premature Withdrawals & Handling of Missing Data

## 10.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | A subject will be considered to have <u>completed study treatment</u> if he/she receives study treatment at Visit 9 (Week 28) and completes the Visit 10/Exit Visit (Week 32). |
| | <ul> <li>A subject will be considered to have <u>completed the study</u> if they continue to participate in the study until the Exit Visit assessments have been completed (regardless of whether the subject completed the study treatment schedule).</li> <li>Subjects who discontinue study treatment or withdraw early will not be replaced</li> </ul> |
| | <ul> <li>in the study.</li> <li>The number of subjects who discontinue study treatment or withdraw early will be summarised and listed.</li> </ul> |
| | All available data from subjects who were withdrawn from the study will be listed and all available data up to and including the date of early withdrawal will be included in summary tables and figures, unless otherwise specified. |
| Pre-Screen Failures, | For the purposes of this study pre-screen failures, screen failures and run-in failures will be defined as follows: |
| Screen<br>Failures<br>and Run-in | <ul> <li>Subjects will be assigned a study number at the time of signing the informed<br/>consent (Pre-screen Visit). Subjects who do not progress to the Screening Visit<br/>will be deemed a <u>pre-screen failure</u>.</li> </ul> |
| Failures | Those subjects that complete at least one additional Visit 1 (Screening) procedure but do not enter the run-in period will be designated as <a href="mailto:screening">screen failures</a> . |
| | Those subjects that enter the run-in but do not subsequently receive study treatment will be designated as <u>run-in failures</u> . |

## 10.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument : |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the listing.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to<br/>be missing data and should be displayed as missing.</li> </ul> |
| | <ul> <li>Results which are found to be below the limit of quantification (BLQ) are not<br/>missing data and will be included in all displays. See Section 10.6 for the<br/>handling of this data.</li> </ul> |
| | The ACQ-5 score will be considered as missing if <4 items of the questionnaire |

| Element | Reporting Detail |
|---|---|
| | are completed at a visit. ACQ-5 Responder/Non-responder category will be missing if the overall ACQ-5 score is missing. |
| | If a blood eosinophil count of zero is reported, it will be imputed with half of the lowest possible blood eosinophil count, where applicable, prior to log transforming the data (Note: this imputation has typically been 0.5 * 0.01 GI/L = 0.005 GI/L for previous mepolizumab studies). |
| | Missing values will not be imputed for any of the other endpoints. |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 10.7.2.1. Handling of Missing or Partial Dates

| Element | Reporting Detail |
|---|---|
| General | The eCRF allows for the possibility of missing or partial dates (i.e., only month and year is captured) to be recorded for event start and end dates. |
| | The recorded missing or partial date will be displayed in listings as captured. |
| Concomitant Medications | Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will<br/>be used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day<br/>(dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| Adverse<br>Events,<br>Exacerbations | <ul> <li>Any partial dates for adverse events and exacerbations will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>However, if these result in a date prior to the start of treatment and the event could possibly have occurred during treatment from the partial information, then the study treatment start date will be assumed to be the start date and hence the event is considered On-treatment (worst case), as per Appendix 4: Treatment Phases.</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The above listed imputations will also be applied when calculating the time to onset and the duration of the event containing missing or partial start and end dates.</li> <li>Start or end dates which are completely missing (i.e. no year specified) will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |

## 10.8. Appendix 8: Values of Potential Clinical Importance

## 10.8.1. Laboratory Values

## **Chemistry Values of Potential Clinical Concern**

| ANALYTE | Age | Sex | SI Units | F3 low | F3 high |
|---|---|---|---|---|---|
| SODIUM | 0+ | Both | MMOL/L | 120 | 160 |
| POTASSIUM | 3+ | Both | MMOL/L | 2.8 | 6.5 |
| CALCIUM | 3+ | Both | MMOL/L | 1.50 | 3.24 |
| PHOSPHORUS,<br>INORG | 3+ | Both | MMOL/L | 0.32 | |
| GLUCOSE | 1+ | Both | MMOL/L | 2.2 | 27.8 |
| ALT (SGPT) | 3-12 | Both | U/L | | >143 (and<br>Total Bilirubin<br>>43) |
| ALT (SGPT) | 13+ | Both | U/L | | >239 (and<br>Total Bilirubin<br>> 43) |

## **Haematology Values of Potential Clinical Concern**

| ANALYTE | Age | Sex | SI Units | F3 low | F3 high |
|---------------------|-----|------|----------|--------|---------|
| HAEMOGLOBIN | 12+ | Both | G/L | 71 | 199 |
| HAEMATOCRIT | 12+ | Both | 1 | 0.201 | 0.599 |
| PLATELET<br>COUNT | 1+ | Both | GI/L | 31 | 1499 |
| WHITE CELL<br>COUNT | 12+ | Both | GI/L | 1.1 | |

## 10.9. Appendix 9: Multicenter Studies

## 10.9.1. Methods for Handling Centres

- In this multicentre global study, enrolment will be presented pooled across investigative sites and countries.
- For the purposes of covariate adjustment in the statistical analysis centres will be grouped into regions. The following regions are defined with consideration for standard of care medical practice, number of subjects enrolled and regulatory considerations:

| Region | Countries |
|----------------|------------------------------------------------------|
| European Union | Belgium, France, Germany, Netherlands, Spain, Sweden |
| Rest of World | Argentina, Canada, United States |

## 10.10. Appendix 10: Examination of Covariates and Subgroups

## 10.10.1. Handling of Covariates

• The following is a list of covariates that will be used in all model-based statistical analyses.

| Category | Subgroups |
|---|---|
| Region | Europe, Rest of World (See Section 10.9 for further details) |
| Exacerbations in the year prior to study (to be included as an ordinal variable) | 2,3,4+ |
| Use of baseline maintenance oral corticosteroids | OCS use, no OCS use |

- Additional covariates of clinical interest may also be considered.
- If the percentage of subjects is small within a particular subgroup, then the subgroup categories may be refined prior to database freeze.
- If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.

## 10.10.2. Handling of Subgroups

The following subgroups are of interest within this study. A separate exploratory analysis of the primary endpoint within each subgroup will be carried out.

Subgroup categories may be further collapsed if there are a small number of subjects in a treatment arm within a subgroup leading to model convergence issues.

The following subgroups are of interest for the primary efficacy endpoint:

- Exacerbations in previous year: <=2, 3, 4+ exacerbations
- Baseline blood eosinophils:  $<150, \ge 150 <300, \ge 300 <500, \ge 500 \text{ cells/}\mu\text{l}$

# 10.11. Appendix 11: Model Checking and Diagnostics for Statistical Analyses

## 10.11.1. Statistical Analysis Assumptions

| Endpoint(s) | Mean change from baseline in ACQ-5 score at Week 32 |
|-------------|-----------------------------------------------------------|
| | Mean change from baseline in SGRQ at Week 32 |
| | Ratio to baseline in blood eosinophil count at Week 32 |
| | Mean change Pre- and Post- bronchodilator FEV1 at Week 32 |
| Analysis | Mixed Model Repeated Measures (MMRM) |

- In the event that this model fails to converge, the list of covariates may be adjusted and/or reduced.
- If there are any important departures from the distributional assumptions, transformations of covariates may be considered or alternative models may be explored as supporting analysis.

| Endpoint(s) | Frequency of exacerbations requiring ED visit/hospitalization during the 32 |
|---|---|
| | <ul> <li>week treatment period</li> <li>Frequency of exacerbations requiring hospitalization during the 32 week treatment period</li> </ul> |
| Analysis | Negative binomial regression analysis |

- In the event that this model fails to converge, the list of covariates may be adjusted and/or reduced.
- Distributional assumptions underlying the model used for analysis will be examined by:
   assessing if a sufficient number of events occurred within covariate categories.
- If there are any important departures from the distributional assumptions, transformations of covariates may be considered or alternative models may be explored as supporting analysis.

## 10.12. Appendix 12: Abbreviations & Trade Marks

## 10.12.1. Abbreviations

| Abbreviation | Description |
|------------------|------------------------------------------------|
| ACQ | Asthma Control Questionnaire |
| ADA | Anti-drug Antibody |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| AIC | Akaike's Information Criteria |
| ALT | Alanine Transaminase |
| ASE | All Subjects Enrolled |
| ATC | Anatomical Therapeutic Chemical |
| BLQ | Below Limit of Quantification |
| BMI | Body Mass Index |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CIL | Clinical Investigation Leader |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Corticosteroid |
| CSR | Clinical Study Report |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| ED | Emergency Department |
| EW | Early Withdrawal |
| FEV <sub>1</sub> | Forced expiratory volume in 1 second |
| FVC | Forced Vital Capacity |
| GCSP | Global Clinical Safety and Pharmacovigilance |
| GSK | GlaxoSmithKline |
| HbsAg | Hepatitis B Surface Antigen |
| ICH | International Conference on Harmonisation |
| ICS | Inhaled Corticosteroids |
| IDSL | Integrated Data Standards Library |
| IG | Implementation Guide |
| IM | Intramuscular |
| IP | Investigational Product |
| IPDISC | Investigational Product Discontinuation |
| IRT | Interactive Response Technology |
| ITT | Intent-To-Treat |
| IV | Intravenous |

| Abbreviation | Description |
|--------------|------------------------------------------------------------|
| LFT | Liver Function Test |
| LLQ | Lower Limit of Quantification |
| MMRM | Mixed Model Repeated Measures |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligram |
| NAb | Neutralising Antibody |
| OCS | Oral Corticosteroids |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PP | Per Protocol |
| PT | Preferred Term |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAMOS NG | Randomization & Medication Ordering System Next Generation |
| RAP | Reporting and Analysis Plan |
| RTF | Rich Text File |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SAS | Statistical Analysis Software |
| SC | Subcutaneous |
| SD | Standard Deviation |
| SDTM | Study Data Tabulation Model |
| SE | Standard Error |
| SGRQ | St. George's Respiratory Questionnaire |
| SMQ | Standard MedDRA Query |
| SOC | System Organ Class |
| SRM | Study Reference Manual |
| TFL | Tables, Figures & Listings |
| TST | Therapeutic Standards Team |
| TSQM | Treatment Satisfaction with Medication Questionnaire |
| VS | Versus/against |

## 10.12.2. Trademarks

| Trader | marks of the GlaxoSmithKline<br>Group of Companies |
|--------|----------------------------------------------------|
| NONE | |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |
| Xolair |

## 10.13. Appendix 13: List of Data Displays

## 10.13.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------|-------------|-------------|
| Study Population | 1.1 to 1.25 | 1.1 |
| Efficacy | 2.1 to 2.46 | 2.1 to 2.11 |
| Safety | 3.1 to 3.56 | 3.1 to 3.2 |
| Section | Listings | |
| ICH and Other Listings | 1 to 44 | |

## 10.13.1.1. Study Population Tables

| Study F | Population: Tab | oles | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable <sup>[1]</sup><br>[Priority] |
| Populat | tion Analysed | | | | |
| 1.1. | ASE | SP1 | Summary of Study Populations | IDSL<br>Include All Subjects Enrolled, Intention<br>to Treat, Per Protocol | SAC |
| Subject | Disposition | | | | |
| 1.2. | ASE | ES6 | Summary of Reasons for Screening and/or Run-In Failures | Journal Requirements | SAC |
| 1.3. | ASE | IE2 | Summary of Failed Inclusion/Exclusion/Continuation Criteria for Screening or Run-in Failures | | SAC |
| 1.4. | ASE | IE2 | Summary of Failed Inclusion/Exclusion/Continuation Criteria for Subjects within the Intent to Treat Population | | SAC |
| 1.5. | ITT | NS1/SHELL | Summary of Number of Subjects by Region, Country and Centre | Add in a column for region, add a total for regions and a total for country EudraCT | SAC |
| 1.6. | ITT | ES1 | Summary of Subject Disposition | ICH E3, GSK CTR, FDAAA, EudraCT | SAC |
| 1.7. | ITT | SD1/SHELL | Summary of Reasons for Withdrawal From Investigational Product | | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.8. | ITT | DM1 | Summary of Demographic Characteristics | ICH E3, GSK CTR, FDAAA, EudraCT | SAC |
| 1.9. | ASE | DM11 | Summary of Age Ranges | EMA, keep row ≥12-17, ≥18-<64, ≥65-<br><84, ≥85 | SAC |
| 1.10. | ITT | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, GSK CTR, FDAAA,<br>EudraCT | SAC |
| 1.11. | ITT | DM6 | Summary of Race and Racial Combination Details | ICH E3, FDA | SAC |

| Study F | opulation: Tab | oles | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable <sup>[1]</sup><br>[Priority] |
| 1.12. | ITT | SHELL | Summary of Asthma History and Baseline Disease Characteristics | Include GERD, CCI, mMRC | SAC |
| 1.13. | ITT | SHELL | Summary of Previous Exacerbation History | | SAC |
| 1.14. | ITT | SU1/SHELL | Summary of History of Tobacco Use | | SAC |
| 1.15. | ITT | SHELL | Summary of Screening and Baseline Lung Function Tests | Include FEV1, FVC, FEV/FVC, %Predicted, Reversibility | SAC |
| Medica | Conditions | | | | |
| 1.16. | ITT | MH4 | Summary of Past Medical Conditions | ICH E3 | SAC |
| 1.17. | ITT | MH4 | Summary of Current Medical Conditions | ICH E3 | SAC |
| 1.18. | ITT | FH1 | Summary of Cardiovascular Assessments – Family History | Note: Family history in women <65 years or men < 55 years (first degree relatives only). Half siblings considered first degree relatives | SAC |
| 1.19. | ITT | FH1 | Summary of Cardiovascular Assessments – Screening Questions | | SAC |
| Prior ar | nd Concomitan | t Medications | | | |
| 1.20. | ITT | SHELL | Summary of Use of Omalizumab Therapy Prior to Treatment | | SAC |

| Study P | Study Population: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable <sup>[1]</sup><br>[Priority] |
| 1.21. | ITT | CM1 | Summary of Asthma Concomitant Medications Started Prior to Treatment by Respiratory Medication Class Group | ICH E3 Footnote: Includes all Asthma medications started before the first dose of investigational product. Multi-component medications displayed under the respiratory medication class of each component Programming note: Display RMC and ingredient as previous Asthma studies | SAC |
| 1.22. | ITT | CM1 | Summary of Asthma Concomitant Medications Taken During Treatment by Respiratory Medication Class Group | Footnote: Multi-component medications displayed under the respiratory medication class of each component Programming note: Display RMC and ingredient as previous Asthma studies | SAC |
| 1.23. | ITT | CM1 | Summary of Asthma Concomitant Medications Taken Post-<br>Treatment by Respiratory Medication Class Group | Footnote: Multi-component medications displayed under the respiratory medication class of each component Programming note: Display RMC and ingredient as previous Asthma studies | SAC |
| 1.24. | ITT | CM1 | Summary of Non-Asthma Medications Taken During Treatment | Footnote: Medications may be displayed under more than one ATC classification | SAC |
| Protoco | ol Deviation | | | | |
| 1.25. | ITT | DV1B | Summary of Protocol Deviations | ICH E3 | SAC |

## 10.13.1.2. Study Population Figures

| Study P | Study Population: Figures | | | | |
|---|---|---|---|---|---|
| No. Population IDSL / TST ID / Example Shell Title Programming Notes Deliveral [Priority | | | | | |
| Subject | Subject Disposition | | | | |
| 1.1 | ITT | SHELL | Time to Subject Withdrawal From Investigation Product | See Study Population Table 1.1<br>(MEA117113 'final' reporting effort),<br>but exclude 'Placebo' and Mepo<br>300mg SC | SAC |

## 10.13.1.3. Efficacy Tables

| Efficacy | r: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Asthma | Control Quest | ionnaire (ACQ-5) | Endpoints | | |
| 2.1. | ITT | SHELL | Summary of Asthma Control Questionnaire (ACQ-5) Score | See Efficacy Table 2.34 (MID200862 'final' reporting effort), but exclude 'Placebo' column Include screening visit in addition to baseline and post-baseline visits | SAC |
| 2.2. | ITT | SHELL | Analysis of Change from Baseline in Asthma Control Questionnaire (ACQ-5) Score Mixed Model Repeated Measures | | SAC |
| 2.3. | PP | SHELL | Sensitivity Analysis of Asthma Control Questionnaire (ACQ-5) Score Responders: Subjects With At Least 0.5-point Improvement from Baseline (Per Protocol Population only) | | SAC |
| 2.4. | ITT | SHELL | Analysis of Change from Baseline in Asthma Control<br>Questionnaire (ACQ-5) by number of exacerbations in previous<br>year | | SAC |
| 2.5. | ITT | SHELL | Analysis of Change from Baseline in Asthma Control Questionnaire (ACQ-5) by baseline blood eosinophils | | SAC |
| 2.6. | ITT | SHELL | Summary of Asthma Control Questionnaire (ACQ-5) Score Responders: Subjects With At Least 0.5-point Improvement from Baseline | See Efficacy Table 2.41 (MID200862 'final' reporting effort), but exclude 'Placebo' column, and rename 'Odd Ratio to Historical Placebo' | SAC |
| St. Geo | rge's Respirato | ory Questionnaire | (SGRQ) Endpoints | | |
| 2.7. | ITT | SHELL | Summary of St George's Respiratory Questionnaire (SGRQ) Total Score | See Efficacy Table 2.01<br>(MID200862 'final' reporting effort),<br>but exclude 'Placebo' column | SAC |

| Efficacy | /: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.8. | ITT | SHELL | Analysis of Change from Baseline in St George's Respiratory<br>Questionnaire (SGRQ) Total Score Mixed Model Repeated<br>Measures | | SAC |
| 2.9. | ITT | SHELL | Summary of St. George's Respiratory Questionnaire (SGRQ)<br>Symptom Domain Score | | SAC |
| 2.10. | ITT | SHELL | Analysis of Change From Baseline in St. George's Respiratory Questionnaire (SGRQ) Symptom Domain Score | | SAC |
| 2.11. | ITT | SHELL | Summary of St. George's Respiratory Questionnaire (SGRQ) Activity Domain Score | | SAC |
| 2.12. | ITT | SHELL | Analysis of Change From Baseline in St. George%'s Respiratory Questionnaire (SGRQ) Activity Domain Score | | SAC |
| 2.13. | ITT | SHELL | Summary of St. George's Respiratory Questionnaire (SGRQ) Impacts Domain Score | | SAC |
| 2.14. | ITT | SHELL | Analysis of Change From Baseline in St. George's Respiratory Questionnaire (SGRQ) Impacts Domain Score | | SAC |
| 2.15. | ITT | SHELL | Summary of St George's Respiratory Questionnaire (SGRQ) Responders: Subjects With At Least 4-point Improvement in Total Score from Baseline | See Efficacy Table 2.24<br>(MID200862 'final' reporting effort),<br>but exclude 'Placebo' column, and<br>rename 'Odd Ratio to Historical<br>Placebo' | SAC |
| Exacerb | oations | | | | |
| 2.16. | ITT | SHELL | Overview of Exacerbations | See Efficacy Table 2.61<br>(MID200862 'final' reporting effort),<br>but exclude 'Placebo' column | SAC |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.17. | ITT | SHELL | Summary of Frequency of Clinically Significant Exacerbations | See Efficacy Table 2.62<br>(MID200862 'final' reporting effort),<br>but exclude 'Placebo' column | SAC |
| 2.18. | ITT | SHELL | Annualised Rate of Clinically Significant Exacerbations | | SAC |
| 2.19. | ITT | SHELL | Analysis of Time to First Clinically Significant Exacerbation | See Efficacy Table 2.68 (MID200862 'final' reporting effort), but exclude 'Placebo' column and Hazard Ration Analysis | SAC |
| 2.20. | ITT | SHELL | Sensitivity Analysis of Annualised Rate of Clinically Significant Exacerbations (on–treatment data only) | | SAC |
| 2.21. | ITT | SHELL | Sensitivity Analysis of Annualised Rate of Clinically Significant Exacerbations (Patients with at least 12 months of prior omalizumab use) | | SAC |
| 2.22. | ITT | SHELL | Summary of Frequency of Exacerbations Requiring Hospitalisation or Emergency Department visits | See Efficacy Table 2.64<br>(MID200862 'final' reporting effort),<br>but exclude 'Placebo' column | SAC |
| 2.23. | ITT | SHELL | Annualised Rate of Exacerbations Requiring Hospitalisation or<br>Emergency Department visits | | SAC |
| 2.24. | ITT | SHELL | Sensitivity Analysis of Annualised Rate of Exacerbations<br>Requiring Hospitalisation or Emergency Department visits (on-<br>treatment data only) | | SAC |
| 2.25. | ITT | SHELL | Summary of Frequency of Exacerbations Requiring Hospitalisation | See Efficacy Table 2.66<br>(MID200862 'final' reporting effort),<br>but exclude 'Placebo' column | SAC |
| 2.26. | ITT | SHELL | Annualised Rate of Exacerbations Requiring Hospitalisation | | SAC |
| Blood E | osinophils | | | | |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.27. | ITT | SHELL | Summary of Blood Eosinophils (109/L) | See Efficacy Table 2.73<br>(MID200862 'final' reporting effort),<br>but exclude 'Placebo' column | SAC |
| 2.28. | ITT | SHELL | Analysis of Change from Baseline in Blood Eosinophils (109/L) | | SAC |
| 2.29. | ITT | SHELL | Analysis of Change from Baseline in Blood Eosinophils (109/L) (on–treatment data only) | | SAC |
| Pre – B | ronchodilator a | and Post – Bronch | odilator FEV1 | | |
| 2.30. | ITT | SHELL | Summary of Clinic Pre-Bronchodilator FEV1 (mL) | See Efficacy Table 2.27<br>(MID200862 'final' reporting effort),<br>but exclude 'Placebo' column | SAC |
| 2.31. | ITT | SHELL | Analysis of Change From Baseline in Clinic Pre-Bronchodilator FEV1 (mL) | See Efficacy Table 2.28<br>(MID200862 'final' reporting effort),<br>but exclude 'Placebo' column and<br>Difference Analysis | SAC |
| 2.32. | ITT | SHELL | Summary of Clinic Post-Bronchodilator FEV1 (mL) | See Efficacy Table 2.49<br>(MID200862 'final' reporting effort),<br>but exclude 'Placebo' column | SAC |
| 2.33. | ITT | SHELL | Analysis of Change From Baseline in Clinic Post-Bronchodilator FEV1 (mL) | See Efficacy Table 2.68<br>(MID200862 'final' reporting effort),<br>but exclude 'Placebo' column and<br>Difference Analysis | SAC |
| Respor | se to Therapy | | | | |
| 2.34. | ITT | SHELL | Summary of Subject Rated Overall Evaluation of Response to Therapy (on–treatment data only) | See Efficacy Table 2.47<br>(MID200862 'final' reporting effort),<br>but exclude 'Placebo' column and<br>Odds Ratio Analysis | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.35. | ITT | SHELL | Summary of Clinician Rated Overall Evaluation of Response to Therapy (on–treatment data only) | | SAC |
| Treatm | ent Satisfacti | on Questionnair | e for Medication (TSQM-9) | | |
| 2.36. | ITT | SHELL | Summary of Treatment Satisfaction Questionnaire for Medication (TSQM – 9) (on–treatment data only) | Summarise the Effectiveness,<br>Convenience and Overall Satisfaction<br>scales separately | SAC |
| Bioma | rkers | | | | |
| 2.37. | ITT | SHELL | Summary of CCL13 (on–treatment data only) | | SAC |
| 2.38. | ITT | SHELL | Summary of CCL17 (on–treatment data only) | | SAC |
| 2.39. | ITT | SHELL | Summary of ECP (on–treatment data only) | | SAC |
| 2.40. | ITT | SHELL | Summary of EDN (on–treatment data only) | | SAC |
| 2.41. | ITT | SHELL | Summary of Eotaxin1 (on–treatment data only) | | SAC |
| 2.42. | ITT | SHELL | Summary of Total IL-5 (on–treatment data only) | | SAC |
| 2.43. | ITT | SHELL | Summary of IL-13 (on–treatment data only) | | SAC |
| 2.44. | ITT | SHELL | Summary of MDC (on–treatment data only) | | SAC |
| 2.45. | ITT | SHELL | Summary of Periostin (on–treatment data only) | | SAC |
| 2.46. | ITT | SHELL | Summary of TSLP (on-treatment data only) | | SAC |

# 10.13.1.4. Efficacy Figures

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Asthma | Control Quest | tionnaire (ACQ-5) | Endpoints | | |
| 2.1. | ITT | SHELL | Figure of Analysis of Asthma Control Questionnaire ( ACQ-5) Score at Each Visit: Mean Change from Baseline | See format of Efficacy Figure 2.11 (MID200862 'final' reporting effort), but exclude 'Placebo' | SAC |
| 2.2. | ITT | SHELL | Cumulative Distribution Function for Change from Baseline in Asthma Control Questionnaire ( ACQ-5) Score at Week 32 | See format of Efficacy Figure 2.14 (MID200862 'final' reporting effort), but exclude 'Placebo' | SAC |
| 2.3. | ITT | SHELL | Figure of Asthma Control Questionnaire (ACQ-5) Responders: Subjects With At Least 0.5-point Improvement in the Score from Baseline | | SAC |
| St. Geo | rge's Respirato | ory Questionnaire | (SGRQ) Endpoints | | |
| 2.4. | ITT | SHELL | Figure of Analysis of St George's Respiratory Questionnaire (SGRQ) Total Score at Each Visit: Mean Change from Baseline | See format of Efficacy Figure 2.01 (MID200862 'final' reporting effort), but exclude 'Placebo' | SAC |
| 2.5. | ITT | SHELL | Figure of St George's Respiratory Questionnaire (SGRQ) Total Score: Change from Baseline At Week 52: Cumulative Distribution Function | See format of Efficacy Figure 2.07 (MID200862 'final' reporting effort), but exclude 'Placebo' | SAC |
| 2.6. | ITT | SHELL | Figure of Analysis of SGRQ by Domain (Mean Change from Baseline at Each Visit) | | SAC |
| 2.7. | ITT | SHELL | Figure of St George's Respiratory Questionnaire (SGRQ) Responders: Subjects With At Least 4-point Improvement in Total Score from Baseline | | SAC |
| Exacer | bations | | | | |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.8. | ITT | SHELL | Kaplan-Meier Cumulative Incidence Curve for Time to First Clinically Significant Exacerbations | See format of Efficacy Figure 2.07 (MID200862 'final' reporting effort), but exclude 'Placebo' | SAC |
| Blood E | osinophils | | | | |
| 2.9. | ITT | SHELL | Figure of Analysis of Blood Eosinophils Ratio Compared to Baseline | See format of Efficacy Figure 6.18 (MEA 115588 'final' reporting effort), but exclude 'Placebo' and mepo 75 mg IV | SAC |
| Pre – bi | ronchodilator a | nd post – bronch | odilator FEV1 | | |
| 2.10. | ITT | SHELL | Figure of Analysis of Pre-Bronchodilator FEV1 (mL) Mean<br>Change From Baseline at Each Visit | See format of Efficacy Figure 2.09 (MID200862 'final' reporting effort), but exclude 'Placebo' | SAC |
| 2.11. | ITT | SHELL | Figure of Analysis of Post-Bronchodilator FEV1 (mL) Mean Change From Baseline at Each Visit | See format of Efficacy Figure 2.09 (MID200862 'final' reporting effort), but exclude 'Placebo' | SAC |

## 10.13.1.5. Safety Tables

| Safety | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Exposu | ire | | | | |
| 3.1 | ITT | SHELL | Summary of Number of Treatments Administered and Time On-<br>Treatment | See format of Study Population Table 1.28 (200862 'final' reporting effort). | SAC |
| Advers | e Events | | | | |
| 3.2 | ITT | SHELL | Overview of All Adverse Events | Add a Total column across all severities | SAC |
| 3.3 | ITT | AE1 | Summary of All On-Treatment Adverse Events by System Organ Class | | SAC |
| 3.4 | ITT | AE5 | Summary of All On-Treatment Adverse Events by System Organ Class and Maximum Intensity | Add a Total column across all severities | SAC |
| 3.5 | ITT | AE1 | Summary of All Post-Treatment Adverse Events by System Organ Class | | SAC |
| 3.6 | ITT | AE5 | Summary of All Post-Treatment Adverse Events by System<br>Organ Class and Maximum Intensity | Add a Total column across all severities | SAC |
| 3.7 | ITT | AE3 | Summary of Common On-Treatment Adverse Events (>=3% in Any Treatment Group) by Overall Frequency | GSK CTR; ≥3% (prior to rounding to nearest percent) | SAC |
| 3.8 | ITT | AE1 | Summary of All On-Treatment Drug-Related Adverse Events by System Organ Class | | SAC |
| 3.9 | ITT | AE5 | Summary of All On-Treatment Drug-Related Adverse Events by System Organ Class and Maximum Intensity | Add a Total column across all severities | SAC |
| 3.10 | ITT | AE1 | Summary of Adverse Events Reported on Day of Dosing by System Organ Class | | SAC |
| 3.11 | ITT | SHELL | Summary of All On-Treatment Adverse Events by Age Group | Add a Total column across all severities | SAC |

| Safety | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.12 | ITT | SHELL | Summary of On-Treatment Adverse Events by Highest Anti Drug Antibody Result At Any Time Post Baseline | | SAC |
| 3.13 | ITT | SHELL | Summary of Post-Treatment Adverse Events by Highest Anti<br>Drug Antibody Result At Any Time Post Baseline | | SAC |
| 3.14 | ITT | AE15 | Summary of Number of Subjects and Occurrences of Common non-Serious Adverse Events by System Organ Class and Preferred Term | GSK CTR; ≥3% (prior to rounding to nearest percent) | SAC |
| Serious | and Other Sig | nificant AEs | | | |
| 3.15 | ITT | AE1 | Summary of Fatal Serious Adverse Events | | SAC |
| 3.16 | ITT | AE1 | Summary of Non-Fatal Serious On-Treatment Adverse Events by System Organ Class | | SAC |
| 3.17 | ITT | AE1 | Summary of Non-Fatal Serious Post-Treatment Adverse Events by System Organ Class | | SAC |
| 3.18 | ITT | AE1 | Summary of Serious Adverse Events by System Organ Class (Pre-Treatment) | | SAC |
| 3.19 | ITT | AE1 | Summary of Serious Adverse Events by System Organ Class (On-Treatment) | | SAC |
| 3.20 | ITT | AE1 | Summary of Serious Adverse Events by System Organ Class (Post-Treatment) | | SAC |
| 3.21 | ITT | AE1 | Summary of Drug-Related Fatal Serious Adverse Events by System Organ Class | | SAC |
| 3.22 | ITT | AE1 | Summary of Drug-Related Serious Adverse Events by System Organ Class and Maximum Intensity | Add a Total column across all severities | SAC |

| Safety | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.23 | ITT | AE3 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by Overall Frequency | | SAC |
| 3.24 | ITT | AE16 | Summary of Number of Subjects and Occurrences of Serious Adverse Events by System Organ Class and Preferred Term | | SAC |
| Advers | e Events of Sp | ecial Interest | | | |
| 3.25 | ITT | AE1 | Summary of AEs meeting Anaphylaxis Criteria (On-Treatment) | Present by Anaphylactic Criterion 1, 2 and 3 rather than SOC as shown in AE1 | SAC |
| 3.26 | ITT | SHELL | Summary Profile of AEs meeting Anaphylaxis Criteria (On-Treatment) | | SAC |
| 3.27 | ITT | AE1 | Summary of AEs Defined by the Investigator as being Systemic (non-allergic or allergic/hypersensitivity) Reactions (On-Treatment) | | SAC |
| 3.28 | ITT | SHELL | Summary Profile of Systemic (non-allergic or allergic/hypersensitivity) Reactions (On-Treatment) | | SAC |
| 3.29 | ITT | SHELL | Summary Profile of Systemic Allergic Reactions (On-Treatment) | | SAC |
| 3.30 | ITT | SHELL | Summary Profile of Systemic Non-Allergic Reactions (On-Treatment) | | SAC |
| 3.31 | ITT | AE1 | Summary of AEs Defined by the Investigator as being Local Injection Site Reactions (On-Treatment) | | SAC |
| 3.32 | ITT | AE1 | Summary of AEs Defined by the Investigator as being Local Injection Site Reactions by Relation to IP (On-Treatment) | | SAC |
| 3.33 | ITT | SHELL | Summary Profile of Local Injection Site Reactions (On-Treatment) | | SAC |

| Safety : | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.34 | ITT | AE3 | Summary of Opportunistic Infections (On-Treatment) | | SAC |
| 3.35 | ITT | SHELL | Summary Profile of Opportunistic Infections (On-Treatment) | | SAC |
| 3.36 | ITT | AE3 | Summary of Malignancies (On-Treatment) | | SAC |
| 3.37 | ITT | SHELL | Summary Profile of Malignancies (On-Treatment) | | SAC |
| 3.38 | ITT | AE1 | Summary of Serious Cardiac, Vascular and Thromboembolic Adverse Events (On-Treatment) | | SAC |
| 3.39 | ITT | SHELL | Summary Profile of Serious Cardiac, Vascular and Thromboembolic Adverse Events (On-Treatment) | | SAC |
| 3.40 | ITT | AE1 | Summary of Serious Ischemic AEs (On-Treatment) | | SAC |
| 3.41 | ITT | SHELL | Summary Profile of Serious Ischemic AEs (On-Treatment) | | SAC |
| 3.42 | ITT | SHELL | Summary of Serious AEs and AEs of Special Interest | See format of Safety Table 7.32 (MEA115588 'final' reporting effort) | SAC |
| Cardiov | ascular Events | 3 | | | • |
| 3.43 | ITT | SHELL | Summary of All Cardiovascular Events Reported by the Investigator | | SAC |
| Labora | tory: Chemistry | 1 | | | |
| 3.44 | ITT | LB1 | Summary of Changes from Baseline in Chemistry Data | Include Baseline values. | SAC |
| 3.45 | ITT | LB3 | Summary of Chemistry Results (Changes from Baseline Relative to the Normal Range) | See also format of Safety Table 7.36 (MEA115588 'final reporting effort) | SAC |
| Labora | tory: Haematol | ogy | | | |
| 3.46 | ITT | LB1 | Summary of Changes From Baseline in Haematology Data | Include Baseline values | SAC |
| 3.47 | ITT | LB3 | Summary of Haematology Results (Changes from Baseline Relative to the Normal Range) | See also format of Safety Table 7.42 (MEA115588 'final reporting effort) | SAC |

| Safety | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Hepato | biliary (Liver) | | | | |
| 3.48 | ITT | LIVER10 | Summary of Subjects Meeting Emergent Hepatobiliary Laboratory Abnormality Criteria | | SAC |
| ECGs | | | | | |
| 3.49 | ITT | EG1 | Summary of ECG Findings | | SAC |
| 3.50 | ITT | EG2 | Summary of Change from Baseline in ECG Values by Visit | Include Baseline values | SAC |
| 3.51 | ITT | SHELL | Summary of Actual and Change From Baseline QTc(F) Values by Category (msec) | | SAC |
| 3.52 | ITT | SHELL | Summary of Actual and Change From Baseline QTc(B) Values by Category (msec) | | |
| Vital Si | gns | | | | |
| 3.53 | ITT | VS1 | Summary of Change From Baseline in Vital Signs by Visit | Include Baseline values | SAC |
| Immun | ogenicity | | | | |
| 3.54 | ITT | SHELL | Summary of ADA Assay Results | See format of Other Assessments<br>Table 8.01 (MEA115588 'final' reporting<br>effort) | SAC |
| 3.55 | ITT | SHELL | Summary of Treatment Emergent ADA Assay Results | | SAC |
| 3.56 | ITT | SHELL | Summary of NAb Assay Results | See format of Other Assessments Table 8.02 (MEA115588 'final' reporting effort) | SAC |

## 10.13.1.6. Safety Figures

| Safety : | Safety : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Laborat | ory | | | | |
| 3.1 | ITT | LIVER9 | Scatter Plot of Maximum Post-Baseline vs. Baseline for ALT | | SAC |
| 3.2 | ITT | LIVER9 | Scatter Plot of Maximum Post-Baseline ALT vs. Maximum Post-Baseline Total Bilirubin | | SAC |

## 10.13.1.7. ICH Listings

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subjec | t Disposition | | | | |
| 1. | ASE | ES7 | Listing of Reasons for Screening Failure or Run-In Failure | | SAC |
| 2. | ASE | IE3 | Listing of Failed Inclusion/Exclusion/Continuation criteria | | SAC |
| 3. | ITT | ES2 | Listing of Reasons for Premature Study Withdrawal | | SAC |
| 4. | ITT | ES2 | Listing of Reasons for Premature Discontinuation of Study Treatment | | SAC |
| Demog | raphics | | | | |
| 5. | ITT | DM2 | Listing of Demographic Characteristics | | SAC |
| 6. | ITT | DM9 | Listing of Race | | SAC |
| Medica | tion Use | | | | |
| 7. | ITT | CM6 | Relationship Between ATC Level 1, Ingredient and Verbatim Text | | SAC |
| Protoc | ol Deviations | | | | |
| 8. | ITT | DV2 | Listing of Important Protocol Deviations | Listing also includes Per-Protocol analysis population exclusions | SAC |
| Efficac | у | | | | |

| ICH Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 9. | ITT | SHELL | Listing of ACQ-5 Data | | SAC |
| 10. | ITT | SHELL | Listing of Exacerbations | See format of Efficacy Listing 6.01 (MEA115588 'final' reporting effort) | SAC |
| Expos | Exposure | | | | |
| 11. | ITT | EX3 | Listing of Exposure Data | | SAC |
| Advers | se Events | | | | |
| 12. | ASE | AE8 | Listing of All Adverse Events | | SAC |
| 13. | ASE | AE7 | Listings of Subject Numbers for Individual Adverse Events | | SAC |
| 14. | ASE | AE2 | Listing of Relationship Between Adverse Event<br>System Organ Classes, Preferred Terms, and<br>Verbatim Text | | SAC |
| Seriou | Serious and Other Significant AEs | | | | |
| 15. | ASE | AE8 | Listing of all Fatal Adverse Events | | SAC |
| 16. | ASE | AE8 | Listing of Non-Fatal Serious Adverse Events | | SAC |
| 17. | ASE | AE14 | Listing of Reasons for Considering as a Serious<br>Adverse Event | | SAC |
| 18. | ITT | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | | SAC |

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Advers | e Events of Sp | pecial Interest | | | |
| 19. | ITT | SHELL | Listing of AEs meeting Anaphylaxis Criteria | See format of Safety Listing 7.10 (MEA115588 'final' reporting effort) | SAC |
| 20. | ITT | SHELL | Listing of Adverse Events Defined by the Investigator as a Systemic (non-allergic or allergic/hypersensitivity) Reaction | See format of Safety Listing 7.07 (MEA115588 'final' reporting effort). Also add a column stating whether AE is related to IP. | SAC |
| 21. | ITT | SHELL | Listing of All Adverse Events Experienced by Subjects with at least one Adverse Event Defined by the Investigator as a Systemic (non-allergic or allergic/hypersensitivity) Reaction | | SAC |
| 22. | ITT | SHELL | Listing of Adverse Events Defined by the Investigator as a Local Injection Site Reaction | See format of Safety Listing 7.09 (MEA115588 'final' reporting effort). Also add a column stating whether AE is related to IP. | SAC |
| 23. | ITT | SHELL | Listing of Opportunistic Infections | See format of Safety Listing 7.10 (MEA115588 'final' reporting effort) | SAC |
| 24. | ITT | SHELL | Listing of Malignancies | See format of Safety Listing 2.03 (mid_mepo_iss 'iss_nda' reporting effort) | SAC |
| 25. | ITT | SHELL | Listing of Serious Cardiac, Vascular and Thromboembolic (CVT) AEs | See format of Safety Listing 7.10 (MEA115588 'final' reporting effort) | SAC |
| 26. | ITT | SHELL | Listing of Serious Ischemic AEs | See format of Safety Listing 7.10 (MEA115588 'final' reporting effort) | SAC |
| Cardiovascular Events | | | | | |

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 27. | ITT | SHELL | Listing of Investigator Reported Cardiovascular Events: Arrhythmias | See format of Safety Listing 7.11 (MEA115588 'final' reporting effort) | SAC |
| 28. | ITT | SHELL | Listing of Investigator Reported Cardiovascular<br>Events: Congestive Heart Failure | See format of Safety Listing 7.12 (MEA115588 'final' reporting effort) | SAC |
| 29. | ITT | SHELL | Listing of Investigator Reported Cardiovascular Events: Cerebrovascular Events/Stroke | See format of Safety Listing 7.13 (MEA115588 'final' reporting effort) | SAC |
| 30. | ITT | SHELL | Listing of Investigator Reported Cardiovascular<br>Events: Deep venous Thrombosis/Pulmonary<br>Embolism | See format of Safety Listing 7.14 (MEA115588 'final' reporting effort) | SAC |
| 31. | ITT | SHELL | Listing of Investigator Reported Cardiovascular<br>Events: Myocardial Infarction/Unstable Angina | See format of Safety Listing 7.15 (MEA115588 'final' reporting effort) | SAC |
| 32. | ITT | SHELL | Listing of Investigator Reported Cardiovascular<br>Events: Peripheral Arterial Thrombosis Embolism | See format of Safety Listing 7.16 (MEA115588 'final' reporting effort) | SAC |
| 33. | ITT | SHELL | Listing of Investigator Reported Cardiovascular<br>Events: Pulmonary Hypertension | See format of Safety Listing 7.17 (MEA115588 'final' reporting effort) | SAC |
| 34. | ITT | SHELL | Listing of Investigator Reported Cardiovascular<br>Events: Revascularisation | See format of Safety Listing 7.18 (MEA115588 'final' reporting effort) | SAC |
| 35. | ITT | SHELL | Listing of Investigator Reported Cardiovascular<br>Events: Valvulopathy | See format of Safety Listing 7.19 (MEA115588 'final' reporting effort) | SAC |
| 36. | ITT | SHELL | Listing of Investigator Reported Cardiovascular<br>Events: All Cause Deaths | See format of Safety Listing 7.20 (MEA115588 'final' reporting effort) | SAC |

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Hepato | Hepatobiliary (Liver) | | | | |
| 37. | ITT | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | | SAC |
| 38. | ITT | LB5 | Chemistry Results for Subjects Meeting Liver<br>Monitoring/Stopping Event Criteria | | SAC |
| 39. | ITT | MH2 | Listing of Medical Conditions for Subjects with Liver<br>Stopping Events | | SAC |
| 40. | ITT | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events | See format of Safety Listing 7.22 (MEA112997 'final' reporting effort) | SAC |
| 41. | ITT | LIVER13 | Listing of Subjects Meeting Hepatobiliary Laboratory Criteria Post-Baseline | | SAC |
| All Lab | All Laboratory | | | | |
| 42. | ITT | LB5 | Listing of Laboratory Data for Subjects with Abnormalities of Potential Clinical Concern | | SAC |
| ECG | ECG | | | | |
| 43. | ITT | EG6 | Listing of ECG Findings for Abnormal Interpretations | | SAC |
| Immunogenicity | | | | | |
| 44. | ITT | SHELL | Listing of Immunogenicity Results | See format of Other Assessments Listing 8.01 (MEA115588 'final' reporting effort) | SAC |

## 10.14. Appendix 14: Example Mock Shells for Data Displays

The data display shells are contained in separate documents which are available on request.